# Statistical Analysis Plan for Final Analysis

Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

A Phase I/II, Randomized, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of MT-2766 in Japanese Adults

| Prepared By: | Mitsubishi Tanabe Pharma Corporation |
|--------------|--------------------------------------|
| Version: | v1.0 |
| Date: | 12Apr2023 |

NCT number: NCT05065619

### APPROVAL FORM

### Statistical Analysis Plan

| Protocol No. | MT-2766-A-101 (CP-PRO-CoVLP-028) |
|---|---|
| Protocol Title | A Phase I/II, Randomized, Placebo-Controlled Study to Evaluate the Safety |
| | and Immunogenicity of MT-2766 in Japanese Adults |
| Version / Date | V3.0 / 16NOV2021 |

### Authors:

| Statistics Author |
|-------------------|
| Print Name: |
| Position: |

### Approved by:

| Statistic Approver | |
|--------------------|------------|
| Print Name: | |
| Position: | |
| Signature: | |
| Approval date: | 2023/04/12 |

### TABLE OF CONTENTS

| 1 Introduction | |
|--------------------------------------------------------|------|
| 2 Study Objective and Endpoints | |
| 2.1 Study Objective(s) | |
| 2.2 Study Endpoint(s) | |
| 2.2.1 Primary Endpoints | 7 |
| 2.2.2 Secondary Endpoints | 7 |
| 2.2.3 Exploratory Endpoints | 8 |
| 3 Study Design | |
| 3.1 Study Phase | 9 |
| 3.2 Study Design | 9 |
| 3.3 Schedule for Tests and Observations | 10 |
| 3.4 Sample Size and Power Considerations | 14 |
| 4 Planned analysis | 15 |
| 4.1 Interim Analysis | 15 |
| 4.2 Final Analysis | 15 |
| 5 Analysis Set | 16 |
| 6 Statistical Considerations | |
| 6.1 Descriptive Statistics | 17 |
| 6.2 Statistical Tests | 17 |
| 7 Data Conventions | 18 |
| 7.1 Analysis Variable Definitions | 18 |
| 7.1.1 Study Subjects | 18 |
| 7.1.1.1 Demographic and Other Baseline Characteristics | 18 |
| 7.1.1.2 Medical History | 18 |
| 7.1.1.3 Prior or Concomitant Medication | |
| 7.1.2 Immunogenicity assessments | 18 |
| 7.1.2.1 Geometric Mean Titer (GMT) | . 18 |
| 7.1.2.2 Geometric Mean Fold Rise (GMFR) | . 19 |
| 7.1.2.3 Seroconversion (SC) Rate | . 19 |
| 7.1.2.4 Immunogenicity values | . 19 |
| 7.1.3 Safety Assessments | . 19 |
| 7.1.3.1 Adverse Events | |
| 7.1.3.2 Laboratory Tests | . 21 |
| 7.2 Analysis Visit Definitions | |
| 7.3 Data Handling Convention for Missing Data | . 22 |
| 8 Statistical Methodology | |
| 8.1 Study Subjects | . 23 |
| 8.1.1 Subject Disposition and Analysis Population | |
| 8.1.2 Demographic and Other Baseline Characteristics | |
| 8.1.3 Medical History | . 23 |
| 8.1.4 Prior or Concomitant Medications | |
| 8.2 Immunogenicity Assessments | . 24 |

| 8.2.1 Primary Immunogenicity Endpoint | . 24 |
|---|---|
| 8.2.1.1 Nab response against the SARS-CoV-2 virus | . 24 |
| 8.2.1.2 Specific Th1 CMI response against the SARS-CoV-2 virus measured by IFN-γ | |
| ELISpot | . 25 |
| 8.2.1.3 Specific Th2 CMI response against the SARS-CoV-2 virus measured by IL-4 | |
| ELISpot | . 25 |
| 8.2.2 Secondary Immunogenicity Endpoints | . 25 |
| 8.2.2.1 Nab response against the SARS-CoV-2 virus | . 25 |
| 8.2.2.2 Specific Th1 CMI response against the SARS-CoV-2 virus measured by IFN-γ | |
| ELISpot | . 26 |
| 8.2.2.3 Specific Th2 CMI response against the SARS-CoV-2 virus measured by IL-4 | |
| ELISpot | . 26 |
| 8.2.2.4 Specific antibody response against the SARS-CoV-2 virus by the total IgG levels | . 26 |
| 8.2.3 Specific CMI response against the SARS-CoV-2 virus measured by the percentage of | of |
| CD4+ T cells expressing functional markers | . 26 |
| 8.2.3.1 Specific antibody response against plant glycans measured by serum IgE levels | . 27 |
| 8.2.4 Other Immunogenicity Endpoints | . 27 |
| 8.2.4.1 The ratio of neutralizing antibody titers: IgG ELISA antibody titers | . 27 |
| 8.3 Safety Assessments | .27 |
| 8.3.1 Primary Safety Endpoint | . 28 |
| 8.3.1.1 The incidences and severity of the solicited AEs | . 28 |
| 8.3.1.2 The incidences, severity, and investigator-assessed causality of unsolicited AEs | . 28 |
| 8.3.1.3 The incidences of serious AEs (SAEs), medically attended AEs (MAAEs), AEs | |
| leading to withdrawal, AEs of special interest (AESIs), and deaths | . 28 |
| 8.3.2 Adverse Events | . 28 |
| 8.3.2.1 Solicited Local and Systemic Adverse Events | . 29 |
| 8.3.2.2 Unsolicited Adverse Events | . 29 |
| 8.3.3 Laboratory Tests | .30 |
| 8.3.4 Vital Signs | 30 |
| 8.3.5 Physical Examinations | 30 |
| 9 Data Presentation Conventions | |
| 9.1 Number of Digits to Report | 31 |
| 9.2 Treatment Groups to Report | 31 |
| 9.3 Analysis Visits to Report | 31 |
| 10 Change from the Protocol | 33 |
| 11 Software | 34 |
| 12 References | 35 |
| Appendix 1 Severity Grades for Solicited Local and Systemic Adverse Events | 36 |
| Appendix 2 VAED | 37 |
| Appendix 3 Hypersensitivity Reactions | 38 |
| Appendix 4 pIMD | |

### **ABBREVIATIONS**

| Abbreviations | Definitions |
|---------------|----------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| ALP | alkaline phosphatase |
| ANCOVA | analysis of covariance |
| AST | aspartate transaminase |
| ATC | anatomical therapeutic chemical |
| BDR | blinded data review |
| BLQ | below limit of quantification |
| BMI | body mass index |
| CI | confidence interval |
| CV | coefficient of variation |
| DP | decimal places |
| DMC | data monitoring committee |
| ECG | electrocardiogram |
| FAS | full analysis set |
| ITT | intent-to-treat |
| LLOQ | lower limit of quantitation |
| MedDRA | medical dictionary for regulatory activities |
| MMRM | mixed model repeated measures |
| PD | pharmacodynamics |
| PDPOP | PD Population |
| PK | pharmacokinetics |
| PKPOP | PK Population |
| PP | per protocol |
| PT | preferred term |
| RAND | all subjects randomized population |
| SAP | statistical analysis plan |
| SAE | serious adverse event |
| SAF | safety population |
| SD | standard deviation |
| SOC | system organ class |
| TEAE | treatment emergent adverse event |
| TESAE | treatment emergent serious adverse events |
| ULN | upper limit of normal range |
| WHO | World Health Organization |

### 1 INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol (v3.0) dated 16-NOV-2021. The plan covers statistical analysis, tabulations and listings of the study data to assess the safety and immunogenicity of MT-2766.

Any statistical analysis details described in this document supersede any description of statistical analysis in the protocol.

### 2 STUDY OBJECTIVE AND ENDPOINTS

### 2.1 Study Objective(s)

The objective of this study is to evaluate the safety and immunogenicity of MT-2766 in Japanese adults.

### 2.2 Study Endpoint(s)

### 2.2.1 Primary Endpoints

The following primary immunogenicity and safety endpoints are for Groups 1 (3.75  $\mu$ g of MT-2766) and Group 2 (placebo for MT-2766 3.75  $\mu$ g).

### Safety:

- 1. The incidences, severity, and investigator-assessed causality of immediate adverse events (AEs) that occur within 30 minutes of first (Day 0) and second (Day 21) injections.
- 2. The incidences and severity of the following solicited AEs that develop within 7 days of first (Day 0) and second (Day 21) injections: (i) local AEs (injection site erythema, injection site swelling, injection site induration, and injection site pain) and (ii) systemic AEs (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck).
- 3. The incidences, severity, and investigator-assessed causality of unsolicited AEs that develop within 21 days of first (Day 0) and second (Day 21) injections.
- 4. The incidences of serious AEs (SAEs), medically attended AEs (MAAEs), AEs leading to withdrawal, AEs of special interest (AESIs), and deaths up to 21 days following first (Day 0) and second (Day 21) injections. AESIs include vaccine-associated enhanced diseases (VAED), hypersensitivity reactions, and potential immune-mediated diseases (pIMDs).

### Immunogenicity:

- 1. SARS-CoV-2 neutralizing antibody (Nab) responses will be analyzed on Days 0, 21, and 42 using the following parameters: geometric mean antibody titer (GMT), seroconversion (SC) rate, and geometric mean fold rise (GMFR);
- 2. SARS-CoV-2-specific T helper 1 (Th1) cell-mediated immune (CMI) responses will be measured on Days 0, 21, and 42 using the interferon (IFN)-γ enzyme-linked immunospot (ELISpot) assay;
- 3. SARS-CoV-2-specific T helper 2 (Th2) CMI responses will be measured on Days 0, 21, and 42 using the interleukin (IL)-4 ELISpot assay.

### 2.2.2 Secondary Endpoints

The following secondary safety and immunogenicity endpoints are for Groups 1 and Group 2.


### Safety:

- 1. The incidences of SAEs, MAAEs, AEs leading to withdrawal, AESIs, and deaths from Day 43 to Day 201:
- 2. The incidences of SAEs, MAAEs, AEs leading to withdrawal, AESIs, and deaths from Day 202 to Day 386;
- 3. The numbers and percentages of subjects with normal and abnormal urine, hematological, and biochemical test results within three days of first (Day 0) and second (Day 21) injections.

### Immunogenicity:

- 1. Persistence of SARS-CoV-2 Nab response will be assessed on Days 128, 201, and 386 using the following parameters: GMT, SC rate, and GMFR.
- 2. SARS-CoV-2-specific antibody responses will be measured on Days 0, 21, and 42 based on the total immunoglobulin G (IgG) level, and the persistence of these antibodies will be analyzed on Days 128, 201, and 386 using the following parameters: GMT, SC rate, and GMFR;
- 3. SARS-CoV-2-specific Th1 CMI responses will be measured on Days 201 and 386 using the IFN-γ ELISpot assay;
- 4. SARS-CoV-2-specific Th2 CMI responses will be measured on Days 201 and 386 using the IL-4 ELISpot assay;

### 2.2.3 Exploratory Endpoints

### Immunogenicity:

- 1. For Group 1 and Group 2, SARS-CoV-2-specific CMI responses will be assessed on Days 0, 21, 42, 201, and 386 based on the percentage of CD4+ T cells expressing functional markers.
- 2. For Group 1 and Group 2, plant glycan-specific antibody responses will be assessed on Days 0, 42, 201 and 386 based on serum IgE levels directed against bromelain-derived cross-reactive carbohydrate determinant MUXF3.
- 3. For Group 1 and Group 2, Further characterization of the MT-2766-induced immune response, if informative;
- 4. For Group 3 (1.875 μg of MT-2766), the same analyses as the primary and secondary endpoints in Groups 1 and Group 2 will be performed as exploratory endpoints.

### Safety

1. For Group 3, the same analyses as the primary and secondary endpoints in Groups 1 and Group 2 will be performed as exploratory endpoints.

### 3 STUDY DESIGN

### 3.1 Study Phase

Study phase: Phase I/II

### 3.2 Study Design

A randomized, multicenter, observer-blinded, placebo-controlled study with Japanese male and female subjects who are seronegative for SARS-COV-2 antibodies and negative for SARS-COV-2 PCR test at screening.

125 subjects will be randomized 4:1 and will receive the same 3.75 µg of MT-2766 or placebo. Subjects will receive two intramuscular (IM) injections 21 days apart on Days 0 and 21, into the deltoid region of the alternating arm (each arm will be injected once), of one of the following blinded treatments:

- Group 1: 3.75 μg of MT-2766 in a final volume of 0.5 mL (n=100)
- Group 2: Placebo for MT-2766 3.75 μg in a final volume of 0.5 mL (n=25)

In addition, subjects in Group 3 (n=20) will receive two IM injections of 1.875  $\mu$ g MT-2766 21 days apart on Days 0 and 21, into the deltoid region of the alternating arm (each arm will be injected once) under open-label. The study may be completed even if fewer than 20 subjects in Group 3 are enrolled.

• Group 3: 1.875 μg of MT-2766 in a final volume of 0.25 mL (n=20)

Subjects will be screened up to 21 days in advance of the first vaccine administration and will demonstrate a satisfactory baseline medical assessment by history, general physical examination, hematological, biochemical, urinalysis and serological analysis. Although tests for SARS-CoV-2 antibodies and PCR will be performed at screening, negative subjects will be enrolled. On Day 0 and Day 21, vaccine administration will occur. Phone contacts will be made after each vaccine administration, specifically for review of the subject's safety and concomitant medication data. Visits to the study site will occur 3 days after each vaccine administration for key safety assessments, and 21 days after each vaccine administration for key safety and immunogenicity assessments.

Subjects will return to the study site on Day 128, Day 201, and Day 386 (3-month, 6-month, and 12-month safety follow-ups and immunogenicity assessments after the last vaccine administration).

In Group 1 and Group 2, the randomization code will be opened after data lock when all subjects in Groups 1 and 2 have reached Day 42. Once the study is unblinded, if the efficacy may be inadequate or unconfirmable, public vaccination will be allowed in Group 1 (3.75 µg of MT-2766). Once the study is unblinded, public vaccination will be allowed in Group 2 (placebo group). In these cases the subject will be withdrawn from the study.

In Group 3, if the efficacy may be inadequate or unconfirmable, public vaccination will be recommended. In this case the subject will be withdrawn from the study.



**Figure 1 Study Flow** 

### 3.3 Schedule for Tests and Observations

Table 1 shows the parameters of tests and observation, and the schedule.

Statistical Analysis Plan for Final Analysis Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

Table 1 Time and Events Schedule

| | Days -21<br>to Day -1 | Day 0 | 0 | Day 1 | Day 3 | Day 8 | Day 15 | Day 21 | 21 | Day 22 | Day 24 | Day 29 | Day 36 | Day 42 | Day49 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (screening) | | - | (+1) | (∓I) | ( <del>±</del> 1) | (±1) | 7#) | (7∓) | (#1) | (#1) | (7∓) | (7#) | (7∓) | (#F) |
| Visit Number | 1 | 7 | | Phone <sup>12</sup> | 3 | Phone <sup>12</sup> | Phone <sup>12</sup> | 7 | 4 | Phone <sup>12</sup> | 5 | Phone <sup>12</sup> | Phone 12 | 9 | Phone 12 |
| | | e - | After<br>vaccin | | | | | Before<br>vaccin | After<br>vaccin | | | | | | |
| | | ation | ation | | | | | ation | ation | | | | | | |
| Informed consent | × | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Medical history /Complications | X | Х | | | | | | | | | | | | | |
| Prior medication | × | Х | | | | | | | | | | | | | į |
| Inclusion/Exclusion criteria | X | Х | | | | | | | | | | | | | |
| Randomization (for Groups 1&2) | | × | | | | | | | | | | | | | |
| Vaccine administration | | X | | | | | | × | ζ. | | | | | | |
| Physical examination | × | × | × | | X | | | × | × | | × | | | × | |
| Vital signs 1 | × | × | Х | | X | | | X | × | | × | | | × | |
| Height(screening only)/Weight/BMI | × | × | | | | | | | | | | | | | |
| SARS-CoV-2 PCR test | × | | | | | | | | | | | | | | |
| SARS-CoV-2 antibody test 2 | × | | | | | | | | | | | | | | |
| Blood chemistry 3/Hematology 4 | × | × | | | × | | | X | | | × | | | × | |
| Urinalysis <sup>5</sup> | × | × | | | X | | | × | | | × | | | × | |
| HIV/HBV/HCV | × | | | | | | | | | | | | | | |
| Pregnancy test 6 | X | X | | | | | | × | | | | | | × | |
| Immunogenicity -Serology (Nab<br>assay/ ELISA/ anti-plant glycans<br>ToF antihodies) 7 | | × | | | | | | × | | | | | | × | |
| Immunogenicity - CMI response (ÆLISvot and ICS) 8 | | × | | | | | | X | | | | | | × | |
| Immediate surveillance | | | × | | | | | | × | | | | | | |
| Provide and collect paper diary and memory aid 9 | | | × | | × | | | Х | | | × | | | х | |
| Collection of solicited local/systemic AEs | | | × | x | х | X | | | X | × | × | × | | | |
| Concomitant medications 10 | | | | | | | | | | | | | | | 1 |
| AEs, SAEs, AESIs, MAAEs " | | | | | | | | | | | | | | | |
| Collection of COVID-19 symptoms | | | Subject<br>vaccina | s will be i<br>tion (Day | nstructed<br>0, post va | Subjects will be instructed to contact the study site if they ext vaccination (Day 0, post vaccination) until the end of the study. | the study<br>until the e | site if t<br>nd of th | hey expe | rience sy | mptoms | of COVID | Subjects will be instructed to contact the study site if they experience symptoms of COVID-19 from the day of the first vaccination (Day 0, post vaccination) until the end of the study. | the day o | f the first |
| | | | | | රි | Confidential | īæ | | | | | | | Page | |

Statistical Analysis Plan for Final Analysis Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

| | Day 77 | Day 105 | Day 12814 | Day 161 | Day 189 | Day 201 | Day 245 | Day 273 | Day 301 | Day 329 | Day 357 | Day 386 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (+14) | (±14) | (±14) | ( <del>+</del> 14) | (±14) | (±14) | (±14) | (±14) | (+14) | (+14) | (±14) | (±14) |
| Visit Number | Phone <sup>12</sup> | Phone 12 | 7 | Phone 12 | Phone 12 | 8 | Phone 12 | Phone <sup>12</sup> | Phone <sup>12</sup> | Phone <sup>12</sup> | Phone <sup>12</sup> | ٥ |
| Informed consent | | | | | | | | | | | | |
| Demographics | | | | | | | | | | | | |
| Medical history /Complications | | | | | | | | | | | | |
| Prior medication | | | | | | | | | | | | |
| Inclusion/Exclusion criteria | | | | | | | | | | | | |
| Randomization | | | | | | | | | | | | |
| Vaccine administration | | | | | | | | | | | | į |
| Physical examination | | | × | | | × | | | | | | × |
| Vital signs 1 | | | × | | | × | | | | | | × |
| Height(screening only)/Weight/BMI | | | | | | | | | | | | |
| SARS-CoV-2 PCR test | | | | | | | | | | | | |
| SARS-CoV-2 antibody test <sup>2</sup> | | | | | | X | | | | | | × |
| Blood chemistry <sup>3</sup> /Hematology <sup>4</sup> | | | | | | | | | | | | |
| Urinalysis 5 | | | | | | | | 111. 111. | | | | |
| HIV/HBV/HCV | | | | | | | | | | | | |
| Pregnancy test 6 | | | X | | | | | | | | | |
| Immunogenicity -Serology (Nabassav/ ELISA/ anti-plant glycans | | | × | | - | × | | | | | | × |
| IgE antibodies)7 | | | | | | | | | | | | |
| Immunogenicity - CMI Response | | | | | | × | | | | | | × |
| Immediate surveillance | | | | | | | | | | | | |
| Provide and collect paper diary and memory aid 9 | | | × | | | × | | | | | | × |
| Collection of solicited | | | | | | | | | | | | |
| local/systemic AEs | į | | | | | | | | | | | 1 |
| Concomitant medications 10 | \<br>\<br>\ | | | | | | | | | | | |
| AES, SAES, AESIS, MAAEs " | • | | | | | | | | | | | A C |
| Collection of COVID-19 symptoms | Subjects will vaccination) | | be instructed to contact the until the end of the study. | et the study a<br>dy. | site if they e | xperience sy | be instructed to contact the study site if they experience symptoms of COVID-19 from the day of the first vaccination (Day 0, post until the end of the study. | 20VID-191 | rom the day | of the first | vaccination ( | Day 0, post |

Biochemistry (serum): Sodium, Potassium, Urea, Creatinine, Glucose, Bilirubin (total), Albumin, Total protein, Alkaline phosphatase, Alamine aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma glutamyl transferase (GGT), Cholesterol (total, HDL, LDL), Triglycerides, Chloride, Calcium, Phosphorus. 1) Resting blood pressure (BP), pulse rate (PR), respiratory rate (RR), and body temperature.
2) Anti-N antibodies will be measured at screening, Days 201 and 386.
3) Biochemistry (serum): Sodium Potessia...


# Statistical Analysis Plan for Final Analysis Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

- Hematology: Hemoglobin, Hematocrit, Red blood cells, Platelets, Mean platelet volume (MPV), Neutrophils, Mean cell hemoglobin (MCH), Mean corpuscular hemoglobin concentration (MCHC), Mean cell volume (MCV), White cell count (total, WBC), Lymphocytes, Monocytes, Eosinophils, Basophils
  - Urinalysis: Macroscopic examination (color, clarity), pH, Specific gravity, Glucose, Protein, Occult blood 3
    - It will be tested in serum at screening and in urine at Days 0, 21, 42, and 128. ම ද
- On Days 21 and 128, the immunogenicity- serology blood sample will be collected for the Nab assay and ELISA only. Anti-plant glycan IgE antibodies will only be measured on Days 0, 42, 201 and 386.
  - Blood samples may not be collected for all subjects.
- If subject cannot use electronic diary, paper diary and memory aid will be acceptable.
- From Day 43, concomitant medication collection will be limited to those used to treat an SAE, medically attended adverse event (MAAE), AE leading to withdrawal, AEs of special interest (AESIs), or an AE that occurred before Day 42 and that is still being used afterwards (i.e. on-going use). 8 6 <u>0</u> 1
  - AEs will be collected up to Day 49; SAEs, MAAEs, AEs leading to withdrawal, and AESIs will be collected through to the end of the study.
    - The study site should contact the subject via the electronic diary, phone, fax or email.
- All efforts will be done to have subjects returning on planned date for Day 21 activities. If for any reason the visit is done before or after this planned date, subsequent visits/procedures will be adjusted accordingly. 13 (2)
- Any subject who withdraws the study will be asked to undergo Day 128 visit procedures within two weeks of withdrawal, if the subject agrees. If a subject is withdrawn from Day 1 to Day 29, solicited local/systemic AEs are including. If a subject is withdrawn from Day 1 to Day 49, unsolicited AEs are investigated. If deemed necessary by (sub)investigator, necessary tests such as biochemistry, hematology, or urinalysis will be performed. 4


### 3.4 Sample Size and Power Considerations

The sample size is not based on a formal statistical power calculation but was considered to be adequate to meet the objectives of the study.

### 4 PLANNED ANALYSIS

### 4.1 Interim Analysis

Interim analyses for immunogenicity and safety will be conducted by MTPC after interim database lock up to Day 42 data in Group 1 and Group 2.

### 4.2 Final Analysis

The database will be locked twice. One is the interim database lock for the above-mentioned interim analyses (see Section 4.1), and the other is the final database lock for the final analyses. The SAP will be finalized and signed off prior to each database lock. Final data analysis will be conducted after the final database lock.

### 5 ANALYSIS SET

The statistical analysis will be based on separate analysis sets, defined as follows:

Safety Analysis Set (SAS):

All subjects who received at least one dose of either the MT-2766 or placebo.

Immunogenicity Intent-to-treat (ITT) Set

All subjects who receive at least one dose of either the MT-2766 or placebo and who have at least 1 post-baseline Immunogenicity assessment.

Immunogenicity Per Protocol (PP) Set

Immunogenicity ITT set who do not have any major protocol violations, and who received either the MT-2766 or placebo. For the Day 21 analysis, this should include the subjects who received the first vaccine dose and had Day 0 and Day 21 immunogenicity sample collections. For the Day 42 analysis, this should include the subjects who received both vaccine doses and had Day 0 and Day 42 immunogenicity sample collections. For the Day 128 analysis, this should include the subjects who received both vaccine doses and had Day 0 and Day 128 immunogenicity sample collections. For the Day 201 analysis, this should include the subjects who received both vaccine doses and had Day 0 and Day 201 immunogenicity sample collections.

All safety analyses will be performed using the SAS. The analyses of all immunogenicity endpoints will be performed using the Immunogenicity PP set as the primary analysis population, and the immunogenicity ITT set, as a secondary analysis population.

### 6 STATISTICAL CONSIDERATIONS

### 6.1 Descriptive Statistics

Unless otherwise specified, continuous data will be summarized descriptively using the number in the analysis set (N), the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. Categorical data will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the treatment group and analysis population being presented, unless otherwise specified.

### 6.2 Statistical Tests

Unless otherwise specified, all formal statistical tests will be done at two-sided significance level of 0.05. Point estimates will be accompanied with two-sided 95% CIs where applicable.

### 7 DATA CONVENTIONS

### 7.1 Analysis Variable Definitions

### 7.1.1 Study Subjects

### 7.1.1.1 Demographic and Other Baseline Characteristics

BMI will be recalculated to 1 decimal place using the following formula:

BMI  $(kg/m^2)$  = weight at screening (kg) /  $\{height at screening (m)\}^2$ 

Significant comorbidities will be defined as co-morbid conditions that puts them at higher risk for severe COVID-19 disease. These significant comorbidities include obesity, hypertension, type 1 or type 2 diabetes, chronic obstructive pulmonary disease (COPD), cardiovascular diseases, chronic kidney diseases, or be immunocompromised persons (e.g., treatment-controlled HIV infection, organ transplant recipients, or patients receiving cancer chemotherapy).

### 7.1.1.2 Medical History

Medical history will be coded according to the MedDRA version 24.1.

### 7.1.1.3 Prior or Concomitant Medication

Medications will be coded according to the WHO Drug Dictionary (WHO-DD) Global B3 version Sep 2021.

### (1) Prior Medication

Prior medication is any medication that was started prior to study vaccine date and ended before study vaccine date.

### (2) Concomitant Medication

Concomitant medication is a medication that starts on or after vaccination date/time at Day 0 or starts before vaccination and is still on-going at the time of the study vaccine.

### 7.1.2 Immunogenicity assessments

### 7.1.2.1 Geometric Mean Titer (GMT)

Continuous immunogenicity endpoints will be logarithmically transformed with 10 as base for analysis. GMT point estimates and the corresponding two-sided 95% CI by treatment group will be calculated as the antilog of the mean and 95% CI of log transformed titer values.

### 7.1.2.2 Geometric Mean Fold Rise (GMFR)

GMFR will be defined as the geometric mean of the ratio of GMTs (Day 21/Day 0, Day 42/Day 0, Day 128/Day 0, Day 201/Day 0).

### 7.1.2.3 Seroconversion (SC) Rate

SC rate is defined as the proportion of subjects achieving SC in the analysis set i.e. subjects with:

- For subjects with detectable Nab/IgG titer at Day 0 (i.e. baseline Nab/IgG titer ≥10):
   a ≥ 4-fold increase in Nab/IgG titers between Day 0 and Day 21/42/128/201,
   respectively.
- For subjects with undetectable Nab/IgG titer at Day 0 (i.e. baseline Nab/IgG titer < 10): Nab/IgG titer of ≥ 40 on Day 21/42/128/201, respectively.

### 7.1.2.4 Immunogenicity values

If antibody titers and concentrations are below the cutoff, i.e the result is of the form '<xx', the value will be set to 0.5\*'xx' before performing GMT calculations. Only samples for which PBMC preparation was performed within 8 hours will be used for analysis.

"Below LOD" in IFN- $\gamma$  and IL-4 data should be considered as "0".

"NR" in IFN-y and IL-4 data should be considered as "not reportable" results.

Value of "< 100" and "IR" in Nab data due to hemolyzed samples should be considered as "not reportable" results.

">ULOQ" in Nab data are results above ULOQ at the maximal dilution and the ">ULOQ" value should be assigned as "64000".

### 7.1.3 Safety Assessments

### 7.1.3.1 Adverse Events

Immediate AEs are defined as any solicited local and systemic AEs and unsolicited AEs occurring within 30 minutes after vaccination. Multiple occurrences of the same event within a subject will be counted once in the maximum severity of symptoms category (potentially life threatening > severe > moderate > mild). Related is defined as AEs with a causality of "Definitely Related", "Probably Related" or "Possibly Related". Not related is defined as AEs with a causality of "Probably Not Related" or "Definitely Not Related".

Adverse events will be coded according to the MedDRA version 24.1.

### (1) Duration of Adverse Events

Duration of Adverse Events (days) = AE stop date – AE start date + 1

### 7.1.3.1.1 Solicited Adverse Events

The PI assessment of a solicited adverse event will always be used when available.

In the event that both an e-diary and a paper diary were completed by the subject for the same solicited AE and the same timepoint, the record with the PI assessment will be used for analysis; otherwise, the paper diary data will be used in the analysis.

Scheduled day and timepoint, if applicable, will be used as record identifier(s) in solicited AE summaries.

### 7.1.3.1.1 Serious Adverse Events (SAE)

An SAE is any untoward medical occurrence (whether or not considered to be related to the study vaccine) that, at any dose:

- Results in death
- Is life-threatening (at the time of the event)
- Requires inpatient hospitalization (≥ 24 hours) or prolongation of existing hospitalization (elective hospitalizations/procedures for pre-existing conditions that have not worsened are excluded)
- Results in persistent or significant disability/incapacity
- Is a congenital abnormality/birth defect

### 7.1.3.1.2 Medically Attended Adverse Events (MAAE)

Medically attended adverse events are defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider.

### 7.1.3.1.3 Adverse Events of Special Interest (AESI)

### 7.1.3.1.3.1 Vaccine Associated Enhanced Disease (VAED)

Safety signal of VAED after exposure to the CoVLP formulation will be closely monitored and assessed by retrieving data for this AESI as follows: AEs within the system organ class (SOC): immune system disorders and high level group term (HLGT): lower respiratory tract disorders (excluding obstruction and infection), cardiac disorders, signs and symptoms not elsewhere classified, vascular disorders, heart failures, arteriosclerosis, stenosis, vascular insufficiency and necrosis, cardiac arrhythmias, myocardial disorders, and vascular hemorrhagic disorders. High level term (HLT): renal failure and impairment and preferred term (PT): pericarditis, coagulopathy, deep vein thrombosis, pulmonary embolism, cerebrovascular accidents, peripheral ischemia, liver injury, Guillain-Barre syndrome, anosmia, ageusia, encephalitis, chilblains, vasculitis, erythema multiforme that require inpatient hospitalization (≥ 24 hours) and have laboratory confirmed SARS-Cov-2 infection will be monitored for assessment of any

potential case of VAED. As this list can be updated during the study, any further changes to the AESI terms will be updated in the Signal Management Plan (SMP).

VAED list is attached in the Appendix.

### 7.1.3.1.3.2 Hypersensitivity Reactions (Anaphylaxis and Severe Allergic Reactions)

All reported events will also be monitored for related hypersensitivity reactions after exposure to the CoVLP formulation. Hypersensitivity will be identified using SMQ broad and narrow terms.

Hypersensitivity reaction list is attached in the Appendix.

### 7.1.3.1.3.3 Potential Immune-Mediated Diseases (pIMD)

Potential immune-mediated diseases (pIMDs) are a subset of AEs associated to the adjuvant that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. pIMDs will be identified using SMQ terms.

pIMD list is attached in the Appendix.

### 7.1.3.2 Laboratory Tests

(1) Laboratory values below the limit of quantification

1/2 LLOQ (lower limit of quantification) will be used for BLQ (below the limit of quantification) data in summary statistics.

### 7.2 Analysis Visit Definitions

The date of the first vaccination is defined as Day 0.

For the Day 21 visits, a window of  $\pm$ 1 days will be applied to sample collection data. For the Day 24 visits, a time window is  $\pm$ 1 days from the date of vaccination 2  $\pm$  3. For the Day 42 visits, a time window is  $\pm$ 2 days from the date of vaccination 2  $\pm$  21. For the Day 128 visits, a time window is  $\pm$ 2 days from the date of vaccination 2  $\pm$  107. For the Day 201 visits, a time window is  $\pm$ 2 days from the date of vaccination 2  $\pm$  180. Subjects who have blood samples for immunogenicity taken outside of the time window for blood sample collection are to be excluded from the IPP set for the specific visit.

Unless otherwise specified, baseline will be the last observed value of the parameter of interest prior to the first vaccination. For post-baseline visit, if there are multiple data in a window, the later data will be used.

### 7.3 Data Handling Convention for Missing Data

### Concomitant medication:

There is no imputation for completely missing dates.

Missing or partial concomitant medication start date:

- If only DAY is missing, use the first day of the month.
- If DAY and Month are both missing, use the first day of the year.

Missing or partial concomitant medication stop date:

- If only DAY is missing, use the last day of the month.
- If DAY and Month are both missing, use the last day of the year.
- If DAY, Month and year are all missing, assign 'continuing' status to stop date.

### Immunogenicity:

Missing immunogenicity data will be retained as missing.

### Adverse events:

There is no imputation for completely missing dates.

Missing or partial AE date:

No imputation of AE partial/missing start/end dates or times will be performed. In case of missing or incomplete AE onset date/time, the AE will be included in the analysis unless the incomplete AE onset date/time information unequivocally indicates that the AE started prior to Day 0.

If an AE allocation to a reporting cannot be unequivocally ascertained due to partial/missing date, the AE will be allocated to all relevant periods.

Missing relatedness and intensity of AEs will not be imputed and will be presented as "Missing".

### Other safety:

For safety summaries, only observed data will be used. Unless otherwise specified, missing safety data will not be imputed.

### 8 STATISTICAL METHODOLOGY

### 8.1 Study Subjects

### 8.1.1 Subject Disposition and Analysis Population

Subject disposition will be presented for all the subjects.

Analysis populations will be summarized on the randomized population.

Randomization details will be listed on the randomized population. Subject disposition will be listed on the randomized population.

Analysis populations will be listed on the randomized population.

### 8.1.2 Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be used.

| | category | descriptive |
|---|---|---|
| Gender | Male, Female | |
| Age(years) | < 65<br>>= 65 | Yes |
| Height(cm) | | Yes |
| Weight(kg) | | Yes |
| BMI(kg/m²) | | Yes |
| Race | Japanese, Other | |
| Ethnicity | Hispanic or Latino, Not<br>Hispanic or Latino | |
| Baseline SARS-<br>CoV-2 antibody<br>test | Positive, Negative | |
| Baseline SARS-<br>CoV-2 PCR test | Positive, Negative | |
| Significant comorbidities | Yes, No | |

Demographic and other baseline characteristics will be summarized on the Immunogenicity ITT set, Immunogenicity PP set and the SAS.

Other baseline characteristics will be listed on the randomized population.

### 8.1.3 Medical History

Medical history will be summarized on the SAS.


Medical history will be listed on the randomized population.

### 8.1.4 Prior or Concomitant Medications

Prior medication and concomitant medication (Up to Day 42 and after Day 43) will be summarized separately on the SAS.

Prior and concomitant medication will be listed on the SAS.

### 8.2 Immunogenicity Assessments

All immunogenicity data will be listed.

The following primary immunogenicity and safety endpoints are for Group 1 and Group 2.

### 8.2.1 Primary Immunogenicity Endpoint

### 8.2.1.1 Nab response against the SARS-CoV-2 virus

The following analyses for the Nab assay will be performed:

- GMT (Day 0, Day 21, and Day 42): The point estimates and the corresponding two-sided 95 % CI by treatment group will be calculated.
- SC rate (Day 21, and Day 42): The point estimates and the corresponding two-sided 95 % CI for subjects achieving SC by treatment group will be calculated.
- GMFR: the geometric mean of the ratio of GMTs (Day 21/Day 0 and Day 42/Day 0) will be calculated.

GMT will be compared between treatment groups using the analysis of variance (ANOVA) model.



For SC rate, Fisher's exact tests will be used to compare between the treatment groups, along with exact Clopper-Pearson 95% CI.

GMFR will be compared using the ANCOVA model. The GMFR will be derived by using ANCOVA to model the difference in the log of the titer values between Day 21 and Day 0 and Confidential


between Day 42 and Day 0, with treatment group as main effect and log-transformed baseline titer as covariate.

The reverse cumulative distribution (RCD) curve (plot % of population against the antibody titres) will be plotted and scatter plot will be created.

# 8.2.1.2 Specific Th1 CMI response against the SARS-CoV-2 virus measured by IFN-γ ELISpot

The specific Th1 CMI response on Day 0, Day 21, and Day 42 measured by IFN- $\gamma$  ELISpot will be compared between treatment groups and timepoints. The Wilcoxon Rank Sum Test, also known as the Mann-Whitney Wilcoxon Test, will be used to estimate the difference in response between treatment groups, along with the corresponding 95% CI for the median and p-value.

Since the response between timepoints are paired data, the Wilcoxon Signed Rank Test will be used to estimate the difference in response between timepoints, along with the corresponding 95% CI for the median and p-value.

Scatter plot of the number of T cells expressing IFN- $\gamma$  will be created.

# 8.2.1.3 Specific Th2 CMI response against the SARS-CoV-2 virus measured by IL-4 ELISpot

The specific Th2 CMI response on Day 0, Day 21, and Day 42 measured by IL-4 ELISpot will be compared between treatment groups and timepoints. The Wilcoxon Rank Sum Test will be used to estimate the difference in response between treatment groups, along with the corresponding 95% CI for the median and p-value.

The Wilcoxon Signed Rank Test will be used to estimate the difference in response between timepoints, along with the corresponding 95% CI for the median and p-value.

Scatter plot of the number of T cells expressing IL-4 will be created.

### 8.2.2 Secondary Immunogenicity Endpoints

### 8.2.2.1 Nab response against the SARS-CoV-2 virus

The following analyses for the Nab assay will be performed:

- GMT (Day 128 and Day 201): The point estimates and the corresponding two-sided 95 % CI by treatment group will be calculated.
- SC rate (Day 128 and Day 201): The point estimates and the corresponding two-sided 95 % CI for subjects achieving SC by treatment group will be calculated.
- GMFR: the geometric mean of the ratio of GMTs (Day 128/Day 0, Day 201/Day 0) will be calculated.

The same methodology as in section 8.2.1.1 will be used.

# 8.2.2.2 Specific Th1 CMI response against the SARS-CoV-2 virus measured by IFN-7 ELISpot

The specific Th1 CMI response induced on Day 201 will be analyzed according to the same methodology as in section 8.2.1.2.

# 8.2.2.3 Specific Th2 CMI response against the SARS-CoV-2 virus measured by IL-4 ELISpot

The specific Th2 CMI response induced on Day 201 will be analyzed according to the same methodology as in section 8.2.1.3.

## 8.2.2.4 Specific antibody response against the SARS-CoV-2 virus by the total IgG levels

The GMT will be calculated on Day 0, Day 21, Day 42 and Day 201 as well as the GMFR (Day 21/Day 0, Day 42/Day 0, Day 201/Day 0). SC rate will be calculated on Day 21, Day 42 and Day 201.

GMT will be compared between treatment groups using the analysis of variance (ANOVA) model.

For SC rate, Fisher's exact test will be used to compare between the treatment groups, along with exact Clopper-Pearson 95% CI.

GMFR will be compared using the ANCOVA model. The GMFR will be derived by using ANCOVA to model the difference in the log of the titer values between Day 21 and Day 0, between Day 42 and Day 0, between Day 201 and Day 0 with treatment group as main effect and log-transformed baseline titer as covariate.

The RCD curve will be plotted.

# 8.2.3 Specific CMI response against the SARS-CoV-2 virus measured by the percentage of CD4+ T cells expressing functional markers

The CMI response on Day 0, Day 21 and Day 42 measured by the percentage of T cells expressing functional markers, using flow cytometry will be compared between treatment groups and timepoints. The Wilcoxon Rank Sum Test will be used to estimate the difference in response between treatment groups, along with the corresponding 95% CI for the median.

The Wilcoxon Signed Rank Test will be used to estimate the difference in response between timepoints, along with the corresponding 95% CI for the median.

### Parameters

CD4+CD8-> IL2+ percent of CD4, CD4+CD8-> IL4+ percent of CD4, CD154+> IFN\_TNF\_IL2\_Poly percent of CD4, CD4+CD8-> IFN\_TNF\_IL2\_Poly percent of CD4

### 8.2.3.1 Specific antibody response against plant glycans measured by serum IgE levels

The specific antibody response against plant glycans induced on Day 0, Day 42 and Day 201 will be analyzed by evaluating the percentage of subjects with detectable IgE levels at each timepoint for each treatment group and the percentage of subjects with undetectable IgE levels at each timepoint for each treatment group along with corresponding two-sided 95% exact (Clopper-Pearson method). The difference in percentage between Day 42 and Day 0, Day 201 and Day 0 and associated 95% CI for the difference will be calculated for each treatment group.

### 8.2.4 Other Immunogenicity Endpoints

### 8.2.4.1 The ratio of neutralizing antibody titers: IgG ELISA antibody titers

The Nab/IgG ratio will be calculated as the antilog of the Nab/IgG ratio and 95 % CI of log transformed titer values. The ratio will be compared between treatment groups using ANOVA.

### 8.3 Safety Assessments

All safety data will be listed.

Safety assessments will be made on the SAS.

Adverse events analyses will be presented for the following reporting period, as applicable:

- <u>Day 0-21 period after vaccination 1:</u> Any AEs meeting the following criteria will be allocated to the first vaccination (vaccination 1) and included in the Day 0-21 analysis for first vaccination:
  - o Any AEs with:
    - onset date/time < date and time of second vaccine administration, if second vaccination is done,
    - else if vaccination 2 not performed, any AEs with onset date ≤ date of vaccination 1+21
- <u>Day 0-21 period after vaccination 2:</u> Any AEs meeting the following criteria will be allocated to second vaccination (vaccination 2) and included in the Day 0-21 analysis for second vaccination:
  - o Any AEs with onset date/time  $\geq$  Date/time of vaccination 2 and with onset date  $\leq$  date of vaccination 2 + 21.

- <u>Day 0-21 period after last vaccination</u>: Any AEs meeting the following criteria will be included in the Day 0-21 period after last vaccination:
  - Any AEs with onset date  $\leq$  date of last vaccination + 21 i.e.:
    - Any AEs with onset date ≤ date of vaccination 2 + 21, if vaccination 2 is performed
  - o Any AEs with onset date  $\leq$  date of vaccination 1 + 21, if vaccination 2 is not performed.

### 8.3.1 Primary Safety Endpoint

### 8.3.1.1 The incidences and severity of the solicited AEs

The incidences and severity of solicited AEs will be summarized by treatment using descriptive statistics.

### 8.3.1.2 The incidences, severity, and investigator-assessed causality of unsolicited AEs

The incidences, severity and relationship of unsolicited AEs will be summarized by treatment using descriptive statistics.

# 8.3.1.3 The incidences of serious AEs (SAEs), medically attended AEs (MAAEs), AEs leading to withdrawal, AEs of special interest (AESIs), and deaths

The incidences of serious AEs (SAEs), medically attended AEs (MAAEs), AEs leading to withdrawal, AEs of special interest (AESIs), and deaths will be summarized by treatment using descriptive statistics.

### 8.3.2 Adverse Events

Overall summary will be conducted through primary safety endpoint.

Overall summary of safety for each Day 0-21 vaccination period:

- Any Immediate AEs (occurring within 30 minutes after vaccination);
  - Immediate solicited AE;
    - Solicited injection site AE
    - Solicited systemic AE
  - Immediate unsolicited AE;
  - Any solicited AE:
    - ≥ Grade 3 Solicited AEs;
    - Solicited Local AEs
    - o Solicited systemic AE;
  - Unsolicited AEs;
    - ≥ Grade 3 unsolicited AEs;
- Serious AEs;
- Related Serious AEs

- Medically Attended AEs;
- Related Medically Attended AEs;
- AEs leading to study withdrawal
- AESI: Overall, VED, Hypersensitivity, potential immune-mediated diseases
- AEs leading to death

Overall summary of safety for up to EOS:

- Unsolicited AEs:
  - Strade 3 unsolicited AEs;
- Serious AEs;
- Related Serious AEs
- Medically Attended AEs;
- Related Medically Attended AEs;
- AEs leading to study withdrawal
- AESI: Overall, VED, Hypersensitivity, potential immune-mediated diseases
- AEs leading to death

### 8.3.2.1 Solicited Local and Systemic Adverse Events

Solicited local and systemic AEs will be summarized through primary safety endpoint for each of the following for overall.

• Solicited local and systemic AEs within first seven days after each vaccination

### 8.3.2.2 Unsolicited Adverse Events

All spontaneous unsolicited AEs will be classified by system organ class (SOC) and preferred term (PT) for each of the following by overall. Unsolicited AEs will be summarized through primary safety endpoint. Most frequent AEs are defined as those that occur > 5% of either of the treatment groups and will only be summarized by PT.

- Most frequent unsolicited AEs
- AESIs
- SAEs
- MAAEs
- AEs leading to death
- AEs leading to withdrawal

### 8.3.3 Laboratory Tests

| Laboratory Test | Parameters |
|---|---|
| Hematology | Haemoglobin, Hematocrit, Red blood cell, Platelets, Mean platelet volume (MPV), White cell count (total, WBC), Neutrophils, Mean cell haemoglobin (MCH), Mean cell concentration (MCHC), Mean cell volume (MCV), Lymphocytes, Monocytes, Eosinophils, Basophils |
| Biochemistry | Sodium, Potassium, Urea, Creatinine, Glucose, Bilirubin (total), Albumin, Total protein, Alkaline phosphatase, Alaninetransferase (ALT), Aspartatetransferase (AST), Gamma glutamyltransferase (GGT), Cholesterol (total, HDL, LDL), Triglyceride, Chloride, Calcium, Phosphorus |
| Urinalysis | Macroscopic examination (color, aspect), pH, Specific gravity, Glucose, Protein, Blood |
| Other | SARS-CoV-2 IgG Antibody, Hepatitis B Virus Surface Antigen, Hepatitis C Virus Antibody |

### 8.3.4 Vital Signs

Absolute values and changes from baseline will be summarized for the following parameters.

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Pulse Rate (beats/min)
- Respiratory Rate (breaths/min)
- Oral Temperature(°C)

### 8.3.5 Physical Examinations

Physical examination will be summarized.

### 9 DATA PRESENTATION CONVENTIONS

### 9.1 Number of Digits to Report

| Statistic | Specification | Apply to |
|---|---|---|
| Minimum, Maximum | Same number of DPs as the data provided in the datasets | All original (i.e. non-derived) |
| | see section 7.3 | All derived data |
| Mean, Median, SD, SE,<br>Confidence intervals | One more DP than above | All |
| Percentages <sup>1</sup> | 1 DP | All |
| Ratios | 3 DPs | A11 |
| p-values <sup>2</sup> | 3 DPs | All |

Percentages: use 1 place beyond the decimal point, except for the following cases: If the percentage is equal to 0, then leave blank, do not use (0) If the percentage is equal to 100, then use "(100)" without a decimal

### 9.2 Treatment Groups to Report

| Treatment Group | For TFLs |
|-----------------|-----------------|
| 3.75 µg MT-2766 | MT-2766 3.75 μg |
| Placebo | Placebo |

### 9.3 Analysis Visits to Report

Immunogenicity:

| Analysis Visit | Apply to |
|---|---|
| Day 0 | All immunogenicity |
| Day 21 | All immunogenicity |
| Day 42 | All immunogenicity |
| Day 128 | All immunogenicity<br>(except for CMI<br>response) |
| Day 201 | All immunogenicity (except for CMI response measured by the percentage of T cells) |

 $<sup>^2</sup>$  p-values: use 3 places beyond the decimal point, except for the following cases: If the p-value is less than 0.001, then use p<0.001

### Safety:

| Analysis Visit | Apply to |
|----------------|----------------------|
| Day 0 | All Laboratory Tests |
| Day 3 | All Laboratory Tests |
| Day 21 | All Laboratory Tests |
| Day 24 | All Laboratory Tests |
| Day 42 | All Laboratory Tests |

| Analysis Visit | Analysis Time | Apply to | |
|----------------|--------------------|-------------|----------------------|
| | Point | Vital Signs | Physical Examination |
| Day 0 | Before vaccination | X | X |
| ***** | After vaccination | X | X |
| Day 3 | | X | X |
| Day 21 | Before vaccination | X | X |
| | After vaccination | X | X |
| Day 24 | | X | X |
| Day 42 | | X | X |
| Day 128 | | X | X |
| Day 201 | | X | X |

Unscheduled visits, retests (same visit number assigned) and follow-up visits will not be displayed in by-visit summary tables, but will be included in the data listings.

Mitsubishi Tanabe Pharma Corporation

### 10 CHANGE FROM THE PROTOCOL

Group 3 was not enrolled. Also, because the study was discontinued, the items on Day 386 and some items were not measured. Only the collected data were included in the tabulation and listings.

Mitsubishi Tanabe Pharma Corporation

### 11 SOFTWARE

All statistical analyses will be performed using SAS version 9.4 or higher.

Statistical Analysis Plan for Final Analysis Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

Mitsubishi Tanabe Pharma Corporation

### 12 REFERENCES

N/A

# APPENDIX 1 SEVERITY GRADES FOR SOLICITED LOCAL AND SYSTEMIC ADVERSE EVENTS

| Symptoms | Severity | | | | |
|---|---|---|---|---|---|
| | None | Grade 1<br>(Mild) | Grade 2<br>(Moderate) | Grade 3<br>(Severe) | Grade 4<br>(Potentially life-<br>threatening) |
| Injection Site Adverse Events (Local Adverse Events) | | | | | |
| Erythema (redness) | < 25 mm | 25 - 50 mm | 51 - 100 mm | > 100 mm | Necrosis or exfoliative dermatitis |
| Swelling | < 25 mm | 25 - 50 mm and<br>does not<br>interfere with<br>activity | 51 – 100 mm or<br>interferes with<br>activity | > 100 mm or<br>prevents daily<br>activity | Necrosis |
| Pain | None | Does not<br>interfere with<br>activity | Repeated use of<br>non-narcotic pain<br>reliever for more<br>than 24 hours or<br>interferes with<br>activity | Any use of<br>narcotic pain<br>reliever or<br>prevents daily<br>activity | Results in a visit<br>to emergency<br>room (ER) or<br>hospitalization |
| Solicited Systemic Ac | lverse Events | | | | |
| Fever (°C or °F) | < 38.0 °C<br>< 100.4 °F | 38.0 - 38.4 °C<br>100.4 - 101.1 °F | 38.5 - 38.9 °C<br>101.2 - 102.0 °F | 39.0 - 40.0 °C<br>102.1 - 104.0 °F | > 40.0 °C<br>> 104.0 °F |
| Headache | None | No interference with activity | Repeated use of<br>non-narcotic pain<br>reliever for more<br>than 24 hours or<br>some interference<br>with activity | Significant; any<br>use of narcotic<br>pain reliever or<br>prevents daily<br>activity | Results in a visit<br>to emergency<br>room (ER) or<br>hospitalization |
| Fatigue | None | No interference with activity | Some interference with activity | Significant;<br>prevents daily<br>activity | Results in a visit<br>to emergency<br>room (ER) or<br>hospitalization |
| Muscle aches | None | No interference with activity | Some interference with activity | Significant;<br>prevents daily<br>activity | Results in a visit<br>to emergency<br>room (ER) or<br>hospitalization |
| Joint aches, chills, feeling of general discomfort or uneasiness (malaise), swelling in the axilla, swelling in the neck | None | No interference with activity | Some interference<br>with activity not<br>requiring medical<br>intervention | Prevents daily<br>activity and<br>requires medical<br>intervention | Results in a visit<br>to emergency<br>room (ER) or<br>hospitalization |
## APPENDIX 2 VAED

| PT | PT Code |
|-----------------------------------------------|----------|
| Asymptomatic COVID-19 | 10084459 |
| Congenital COVID-19 | 10085080 |
| Coronavirus infection | 10051905 |
| Coronavirus pneumonia | 10084381 |
| Coronavirus test positive | 10070255 |
| COVID-19 | 10084268 |
| COVID-19 immunisation | 10084457 |
| COVID-19 pneumonia | 10084380 |
| COVID-19 prophylaxis | 10084458 |
| COVID-19 treatment | 10084460 |
| Exposure to SARS-CoV-2 | 10084456 |
| Multisystem inflammatory syndrome | 10086091 |
| Multisystem inflammatory syndrome in adults | 10085850 |
| Multisystem inflammatory syndrome in children | 10084767 |
| Occupational exposure to SARS-CoV-2 | 10084394 |
| Post-acute COVID-19 syndrome | 10085503 |
| SARS-CoV-2 antibody test positive | 10084491 |
| SARS-CoV-2 carrier | 10084461 |
| SARS-CoV-2 RNA decreased | 10085496 |
| SARS-CoV-2 RNA fluctuation | 10085497 |
| SARS-CoV-2 RNA increased | 10085495 |
| SARS-CoV-2 sepsis | 10084639 |
| SARS-CoV-2 test false negative | 10084480 |
| SARS-CoV-2 test positive | 10084271 |
| SARS-CoV-2 viraemia | 10084640 |
| Suspected COVID-19 | 10084451 |
| Thrombosis with thrombocytopenia syndrome | 10086158 |
| Vaccine derived SARS-CoV-2 infection | 10085492 |

# APPENDIX 3 HYPERSENSITIVITY REACTIONS

| PT | PT Code |
|--------------------------------------------|----------|
| Acquired C1 inhibitor deficiency | 10081035 |
| Acute generalised exanthematous pustulosis | 10048799 |
| Administration related reaction | 10069773 |
| Administration site dermatitis | 10075096 |
| Administration site eczema | 10075099 |
| Administration site hypersensitivity | 10075102 |
| Administration site rash | 10071156 |
| Administration site recall reaction | 10075964 |
| Administration site urticaria | 10075109 |
| Administration site vasculitis | 10075969 |
| Allergic bronchitis | 10052613 |
| Allergic colitis | 10059447 |
| Allergic cough | 10053779 |
| Allergic cystitis | 10051394 |
| Allergic eosinophilia | 10075185 |
| Allergic gastroenteritis | 10075308 |
| Allergic hepatitis | 10071198 |
| Allergic keratitis | 10057380 |
| Allergic lymphangitis | 10086007 |
| Allergic oedema | 10060934 |
| Allergic otitis externa | 10075072 |
| Allergic otitis media | 10061557 |
| Allergic pharyngitis | 10050639 |
| Allergic reaction to excipient | 10078853 |
| Allergic respiratory disease | 10063532 |
| Allergic respiratory symptom | 10063527 |
| Allergic sinusitis | 10049153 |
| Allergic stomatitis | 10079554 |
| Allergic transfusion reaction | 10066173 |
| Allergy alert test positive | 10075479 |
| Allergy test positive | 10056352 |
| Allergy to immunoglobulin therapy | 10074079 |
| Allergy to surgical sutures | 10077279 |
| Allergy to vaccine | 10055048 |
| Anal eczema | 10078682 |
| Anaphylactic reaction | 10002198 |
| Anaphylactic shock | 10002199 |
| Anaphylactic transfusion reaction | 10067113 |

| | 110000016 |
|----------------------------------------------------------|-----------|
| Anaphylactoid reaction | 10002216 |
| Anaphylactoid shock | 10063119 |
| Anaphylaxis treatment | 10002222 |
| Angioedema | 10002424 |
| Antiallergic therapy | 10064059 |
| Antiendomysial antibody positive | 10065514 |
| Anti-neutrophil cytoplasmic antibody positive vasculitis | 10050894 |
| Application site dermatitis | 10003036 |
| Application site eczema | 10050099 |
| Application site hypersensitivity | 10063683 |
| Application site rash | 10003054 |
| Application site recall reaction | 10076024 |
| Application site urticaria | 10050104 |
| Application site vasculitis | 10076027 |
| Arthritis allergic | 10061430 |
| Aspirin-exacerbated respiratory disease | 10075084 |
| Atopic cough | 10081492 |
| Atopy | 10003645 |
| Blepharitis allergic | 10005149 |
| Blood immunoglobulin E abnormal | 10005589 |
| Blood immunoglobulin E increased | 10005591 |
| Bromoderma | 10006404 |
| Bronchospasm | 10006482 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Catheter site dermatitis | 10073992 |
| Catheter site eczema | 10073995 |
| Catheter site hypersensitivity | 10073998 |
| Catheter site rash | 10052271 |
| Catheter site urticaria | 10052272 |
| Catheter site vasculitis | 10074014 |
| Chronic eosinophilic rhinosinusitis | 10071399 |
| Chronic hyperplastic eosinophilic sinusitis | 10071380 |
| Circulatory collapse | 10009192 |
| Circumoral oedema | 10052250 |
| Circumoral swelling | 10081703 |
| Conjunctival oedema | 10010726 |
| Conjunctivitis allergic | 10010744 |
| Contact stomatitis | 10067510 |
| Contrast media allergy | 10066973 |
| Contrast media reaction | 10010836 |

| | 1 |
|-------------------------------------------------------|----------|
| Corneal oedema | 10011033 |
| Cross sensitivity reaction | 10011411 |
| Cutaneous vasculitis | 10011686 |
| Dennie-Morgan fold | 10062918 |
| Dermatitis | 10012431 |
| Dermatitis acneiform | 10012432 |
| Dermatitis allergic | 10012434 |
| Dermatitis atopic | 10012438 |
| Dermatitis bullous | 10012441 |
| Dermatitis contact | 10012442 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Dermatitis herpetiformis | 10012468 |
| Dermatitis infected | 10012470 |
| Dermatitis psoriasiform | 10058675 |
| Device allergy | 10072867 |
| Dialysis membrane reaction | 10076665 |
| Distributive shock | 10070559 |
| Documented hypersensitivity to administered | |
| product | 10076470 |
| Drug eruption | 10013687 |
| Drug hypersensitivity | 10013700 |
| Drug provocation test | 10074350 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Eczema | 10014184 |
| Eczema infantile | 10014198 |
| Eczema nummular | 10014201 |
| Eczema vaccinatum | 10066042 |
| Eczema vesicular | 10058681 |
| Eczema weeping | 10055182 |
| Encephalitis allergic | 10056387 |
| Encephalopathy allergic | 10014627 |
| Eosinophilic granulomatosis with polyangiitis | 10078117 |
| Epidermal necrosis | 10059284 |
| Epidermal necrosis Epidermolysis | 10053177 |
| Epidermolysis Epidermolysis bullosa | 10033177 |
| | 10014989 |
| Epiglottic oedema Erythema multiforme | 10015029 |
| | 10013218 |
| Erythema nodosum | 10013228 |
| Exfoliative rash | 10004379 |

| Eye allergy | 10015907 |
|--------------------------------------------|----------|
| Eye oedema | 10052139 |
| Eye swelling | 10032133 |
| Eyelid oedema | 10015993 |
| Face oedema | 10016029 |
| Fixed eruption | 10016741 |
| Generalised bullous fixed drug eruption | 10084905 |
| Giant papillary conjunctivitis | 10018258 |
| Gingival oedema | 10049305 |
| Gingival swelling | 10049303 |
| Gleich's syndrome | 10016231 |
| Haemorrhagic urticaria | 10059499 |
| Hand dermatitis | 10058898 |
| | 10038838 |
| Henoch-Schonlein purpura | 10019017 |
| Henoch-Schonlein purpura nephritis | 10069440 |
| Heparin-induced thrombocytopenia | 10062306 |
| Hypersensitivity | 10020731 |
| Hypersensitivity myocarditis | 10081004 |
| Hypersensitivity pneumonitis | 10081988 |
| Hypersensitivity vasculitis | |
| Idiopathic urticaria | 10021247 |
| Immediate post-injection reaction | |
| Immune thrombocytopenia | 10083842 |
| Immune tolerance induction | 10070581 |
| Implant site dermatitis | 10063855 |
| Implant site hypersensitivity | 10063858 |
| Implant site rash | 10063786 |
| Implant site urticaria | 10063787 |
| Incision site dermatitis | 10073168 |
| Incision site rash | 10073411 |
| Infusion related hypersensitivity reaction | 10082742 |
| Infusion related reaction | 10051792 |
| Infusion site dermatitis | 10065458 |
| Infusion site eczema | 10074850 |
| Infusion site hypersensitivity | 10065471 |
| Infusion site rash | 10059830 |
| Infusion site recall reaction | 10076085 |
| Infusion site urticaria | 10065490 |
| Infusion site vasculitis | 10074851 |
| Injection related reaction | 10071152 |
| Injection site dermatitis | 10022056 |

| Injection site eczema1006622Injection site hypersensitivity1002207Injection site rash1002209Injection site recall reaction1006679 |
|---|
| Injection site rash 1002209 |
| Injection site recall reaction 1006679 |
| Injection site urticaria 1002210 |
| Injection site vasculitis 1006799 |
| Instillation site hypersensitivity 1007361 |
| Instillation site rash 1007362 |
| Instillation site urticaria 1007362 |
| Interstitial granulomatous dermatitis 1006797 |
| Intestinal angioedema 1007622 |
| Iodine allergy 1005209 |
| Kounis syndrome 1006916 |
| Laryngeal oedema 1002384 |
| Laryngitis allergic 1006486 |
| Laryngospasm 1002389 |
| Laryngotracheal oedema 1002389 |
| Limbal swelling 1007049 |
| Lip oedema 1002455 |
| Lip swelling 1002457 |
| Mast cell activation syndrome 1007521 |
| Mast cell degranulation present 1007660 |
| Medical device site dermatitis 1007557 |
| Medical device site eczema 1007557 |
| Medical device site hypersensitivity 1007557 |
| Medical device site rash 1007558 |
| Medical device site recall reaction 1007614 |
| Medical device site urticaria 1007558 |
| Mouth swelling 1007520 |
| Mucocutaneous rash 1005667 |
| Multiple allergies 1002816 |
| Nephritis allergic 1002912 |
| Nikolsky's sign 1002941 |
| Nodular rash 1007580 |
| Nutritional supplement allergy 1008404 |
| Oculomucocutaneous syndrome 1003008 |
| Oculorespiratory syndrome 100673 |
| Oedema mouth 100301 |
| Oral allergy syndrome 1006835 |
| Oropharyngeal blistering 1006795 |
| Oropharyngeal oedema 1007878 |

| Oropharyngeal swelling Palatal oedema Palatal swelling Palisaded neutrophilic granulomatous dermatitis Palpable purpura Pathergy reaction Perioral dermatitis Periorbital oedema Periorbital swelling Pharyngeal oedema Pharyngeal swelling Polymers allergy Procedural shock Pruritus allergic 100 1 | 0031111<br>0031118<br>0056998<br>0074403<br>0068809<br>0056872<br>0074332<br>0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347 |
|---|---|
| Palatal oedema 10 Palatal swelling 10 Palisaded neutrophilic granulomatous dermatitis 10 Palpable purpura 10 Pathergy reaction 10 Perioral dermatitis 10 Periorbital oedema 10 Periorbital swelling 10 Pharyngeal oedema 10 Pharyngeal swelling 10 Pharyngeal swelling 10 Procedural shock 10 Pruritus allergic 10 | 0056998<br>0074403<br>0068809<br>0056872<br>0074332<br>0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Palatal swelling Palisaded neutrophilic granulomatous dermatitis Palpable purpura 10 Pathergy reaction Perioral dermatitis 11 Periorbital oedema 12 Periorbital swelling Pharyngeal oedema 13 Pharyngeal swelling Polymers allergy Procedural shock Pruritus allergic 16 17 18 19 10 | 0074403<br>0068809<br>0056872<br>0074332<br>0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894 |
| Palisaded neutrophilic granulomatous dermatitis Palpable purpura Pathergy reaction Perioral dermatitis Periorbital oedema Periorbital swelling Pharyngeal oedema Pharyngeal swelling Polymers allergy Procedural shock Pruritus allergic | 0068809<br>0056872<br>0074332<br>0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Palpable purpura 10 Pathergy reaction 10 Perioral dermatitis 10 Periorbital oedema 10 Periorbital swelling 10 Pharyngeal oedema 10 Pharyngeal swelling 10 Pharyngeal swelling 10 Procedural shock 10 Pruritus allergic 10 | 0056872<br>0074332<br>0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Pathergy reaction 10 Perioral dermatitis 10 Periorbital oedema 10 Periorbital swelling 10 Pharyngeal oedema 10 Pharyngeal swelling 10 Pharyngeal swelling 10 Procedural shock 10 Pruritus allergic 10 | 0074332<br>0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Perioral dermatitis Periorbital oedema Periorbital swelling Pharyngeal oedema Pharyngeal swelling Polymers allergy Procedural shock Pruritus allergic 10 1 | 0034541<br>0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Periorbital oedema 10 Periorbital swelling 10 Pharyngeal oedema 10 Pharyngeal swelling 10 Pharyngeal swelling 10 Polymers allergy 10 Procedural shock 10 Pruritus allergic 10 | 0034545<br>0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Periorbital swelling Pharyngeal oedema Pharyngeal swelling Polymers allergy Procedural shock Pruritus allergic 10 1 | 0056647<br>0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Pharyngeal oedema 10 Pharyngeal swelling 10 Polymers allergy 10 Procedural shock 10 Pruritus allergic 10 | 0034829<br>0082270<br>0086347<br>0080894<br>0063438 |
| Pharyngeal swelling Polymers allergy 10 Procedural shock 11 Pruritus allergic 11 | 0082270<br>0086347<br>0080894<br>0063438 |
| Polymers allergy 10 Procedural shock 10 Pruritus allergic 10 | 0086347 |
| Procedural shock 10 Pruritus allergic 10 | 0080894 |
| Pruritus allergic 10 | 0063438 |
| Radioallergosorbent test positive 10 | 0037789 |
| Rash 10 | 0037844 |
| Rash erythematous 10 | 0037855 |
| Rash follicular 16 | 0037857 |
| Rash macular 10 | 0037867 |
| Rash maculo-papular 10 | 0037868 |
| Rash maculovesicular 10 | 0050004 |
| Rash morbilliform 10 | 0037870 |
| Rash neonatal 10 | 0037871 |
| Rash papulosquamous 10 | 0037879 |
| Rash pruritic 10 | 0037884 |
| Rash pustular 10 | 0037888 |
| Rash rubelliform 10 | 0057984 |
| Rash scarlatiniform 10 | 0037890 |
| Rash vesicular 10 | 0037898 |
| Reaction to azo-dyes 10 | 0037973 |
| Reaction to colouring 10 | 0037974 |
| Reaction to excipient 10 | 0079925 |
| Reaction to food additive 1 | 0037977 |
| Reaction to preservatives 1 | 0064788 |
| Red man syndrome 1 | 0038192 |
| Rhinitis allergic 1 | 0039085 |
| Scleral oedema 1 | 0057431 |
| Scleritis allergic 1 | 0051126 |
| Scrotal dermatitis 1 | 0083260 |
| Scrotal oedema 1 | 0039755 |

| Serum sickness-like reaction 10040402 | Serum sickness | 10040400 |
|---|---|---|
| Shock 10040560 Shock symptom 10040581 SJS-TEN overlap 10083164 Skin necrosis 10040893 Skin reaction 10040914 Skin test positive 10040934 Solar urticaria 10041307 Solvent sensitivity 10041316 Stevens-Johnson syndrome 10042033 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10043967 Toxic epidermal necrolysis 10043967 Toxic epidermal necrolysis 10043967 Toxic skin eruption 10057970 Tracheal oedema 10044223 Type I hypersensitivity 10045240 Type II hypersensitivity 10045240 Type III immune complex mediated reaction 10053613 Urticaria 10046735 Urticaria chronic 10053613 Urticaria papular 10046742 Urticaria pigmentosa <th< td=""><td></td><td></td></th<> | | |
| Shock symptom 10040581 SIS-TEN overlap 10083164 Skin necrosis 10040893 Skin reaction 10040914 Skin test positive 10040934 Solar urticaria 10041307 Solvent sensitivity 10041316 Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swellen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type II hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046770 Urt | | |
| SIS-TEN overlap 10083164 Skin necrosis 10040893 Skin reaction 10040914 Skin test positive 10040934 Solar urticaria 10041307 Solvent sensitivity 10041316 Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic epidermal necrolysis 10044223 Toxic epidermal necrolysis 10044223 Type I hypersensitivity 10044296 Type II hypersensitivity 10044296 Type II hypersensitivity 10054000 Type IV hypersensitivity reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria chlonic 10053613 Urticaria contact 10046740 | | |
| Skin necrosis 10040893 Skin reaction 10040914 Skin test positive 10040934 Solar urticaria 10041307 Solvent sensitivity 10041316 Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044226 Type I hypersensitivity 10045240 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046740 Urticaria cholinergic 10046740 Urticaria papular 10046742 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046752 Urt | | |
| Skin reaction 10040914 Skin test positive 10040934 Solar urticaria 10041307 Solvent sensitivity 10041316 Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III hypersensitivity 10054000 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria pipular 10046740 Urticaria pipular 10046751 Urticaria pigmentosa 10046752 Urticarial dermatitis 10046752 Urticarial ves | | |
| Skin test positive 10040934 Solar urticaria 10041307 Solvent sensitivity 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type II hypersensitivity 10054000 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria papular 10046750 Urticaria pigmentosa 10046750 Urticaria pigmentosa 10046751 Urticarial dermatitis 1004820 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069487 Va | | |
| Solar urticaria 10041307 Solvent sensitivity 10042033 Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type II hypersensitivity 10054000 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticaria pigmentosa 10046751 Urticarial dermatitis 1004820 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069489 | | |
| Solvent sensitivity 10041316 Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticarial dermatitis 10046752 Urticarial dermatitis 10046755 Urticarial vasculitis 10069477 Vaccination site dermatitis 10069489 </td <td></td> <td></td> | | |
| Stevens-Johnson syndrome 10042033 Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10033613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticarial dermatitis 10082290 Urticarial vasculitis 10048220 Vaccination site dermatitis 10069477 Vaccination site exfoliation 10068880 | | |
| Stoma site hypersensitivity 10074509 Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria chronic 10052568 Urticaria papular 10046740 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10069477 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10068880 | | |
| Stoma site rash 10059071 Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | |
| Swelling face 10042682 Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 1004820 Vaccination site dermatitis 10076161 Vaccination site hypersensitivity 10068880 | | _ |
| Swelling of eyelid 10042690 Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria chronic 10046740 Urticaria chronic 10046740 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site eczema 10076161 Vaccination site hypersensitivity 10068880 | | |
| Swollen tongue 10042727 Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type III hypersensitivity 10054000 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046735 Urticaria chronic 10052568 Urticaria papular 10046742 Urticaria physical 10046750 Urticaria vesiculosa 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site eczema 10076161 Vaccination site hypersensitivity 10068880 | | |
| Symmetrical drug-related intertriginous and flexural exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type III impure complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site hypersensitivity 10068880 | | |
| exanthema 10078325 Tongue oedema 10043967 Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria chloinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10046755 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10042727 |
| Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type II hypersensitivity 10045240 Type III hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria pigmentosa 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048220 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10078325 |
| Toxic epidermal necrolysis 10044223 Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048220 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | Tongue oedema | 10043967 |
| Toxic skin eruption 10057970 Tracheal oedema 10044296 Type I hypersensitivity 10054000 Type III hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria vesiculosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10044223 |
| Tracheal oedema 10044296 Type I hypersensitivity 10045240 Type III hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10057970 |
| Type II hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10044296 |
| Type II hypersensitivity 10054000 Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | Type I hypersensitivity | 10045240 |
| Type III immune complex mediated reaction 10053614 Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10054000 |
| Type IV hypersensitivity reaction 10053613 Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | Type III immune complex mediated reaction | 10053614 |
| Urticaria 10046735 Urticaria cholinergic 10046740 Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10053613 |
| Urticaria chronic 10052568 Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10046735 |
| Urticaria contact 10046742 Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site excema 10076161 Vaccination site hypersensitivity 10068880 | Urticaria cholinergic | 10046740 |
| Urticaria papular 10046750 Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site eczema 10076161 Vaccination site hypersensitivity 10068880 | Urticaria chronic | 10052568 |
| Urticaria physical 10046751 Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site eczema 10076161 Vaccination site hypersensitivity 10068880 | Urticaria contact | 10046742 |
| Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site eczema 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | Urticaria papular | 10046750 |
| Urticaria pigmentosa 10046752 Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site eczema 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10046751 |
| Urticaria vesiculosa 10046755 Urticarial dermatitis 10082290 Urticarial vasculitis 10048820 Vaccination site dermatitis 10069477 Vaccination site eczema 10076161 Vaccination site exfoliation 10069489 Vaccination site hypersensitivity 10068880 | | 10046752 |
| Urticarial vasculitis10048820Vaccination site dermatitis10069477Vaccination site eczema10076161Vaccination site exfoliation10069489Vaccination site hypersensitivity10068880 | | 10046755 |
| Vaccination site dermatitis10069477Vaccination site eczema10076161Vaccination site exfoliation10069489Vaccination site hypersensitivity10068880 | Urticarial dermatitis | 10082290 |
| Vaccination site eczema10076161Vaccination site exfoliation10069489Vaccination site hypersensitivity10068880 | Urticarial vasculitis | 10048820 |
| Vaccination site eczema10076161Vaccination site exfoliation10069489Vaccination site hypersensitivity10068880 | Vaccination site dermatitis | 10069477 |
| Vaccination site exfoliation10069489Vaccination site hypersensitivity10068880 | | 10076161 |
| Vaccination site hypersensitivity 10068880 | Vaccination site exfoliation | 10069489 |
| | | 10068880 |
| | | 10069482 |

| Vaccination site recall reaction 10076188 Vaccination site urticaria 10069622 Vaccination site vasculitis 10076191 Vaccination site vesicles 10069623 Vaginal ulceration 10046943 Vascular access site dermatitis 10085938 Vascular access site ezema 10085939 Vasculitic rash 10047111 Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 1006273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Allergy to chemicals 10061626 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10061425 Anti-insulin antibody increased 10061427 Anti-insulin receptor antibo | · | |
|---|---|---|
| Vaccination site vasculitis 10076191 Vaccination site vesicles 10069623 Vaginal ulceration 10046943 Vascular access site dermatitis 10085938 Vasculitic rash 10047111 Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075289 Allergy to chemicals 10061626 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10061425 Antibody test abnormal 10061425 Anti-insulin antibody increased 10053814 Anti-insulin antibody positive 10063814 Anti-insulin r | Vaccination site recall reaction | 10076188 |
| Vaccination site vesicles 10069623 Vaginal ulceration 10046943 Vascular access site dermatitis 10085938 Vascular access site eczema 10085939 Vasculitic rash 10047111 Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 1006273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginitis allergic 10080783 Acute respiratory failure 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10061426 Anti-insulin antibody increased 10053814 Anti-insulin antibody positive 100633814 Anti-insulin receptor antibody increased 10068226 Application site photosensitivity reaction 10058730 | Vaccination site urticaria | 10069622 |
| Vaginal ulceration 10046943 Vascular access site dermatitis 10085938 Vasculitic rash 10047111 Vernal keratoconjunctivitis 10047111 Vernal keratoconjunctivitis 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 1001889 Antibody test abnormal 10061425 Anti-insulin antibody increased 100533815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody positive 10068226 Application site photosensitivity reaction 10058730 <t< td=""><td>Vaccination site vasculitis</td><td></td></t<> | Vaccination site vasculitis | |
| Vascular access site dermatitis 10085938 Vascular access site eczema 10085939 Vasculitic rash 10047111 Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10061626 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody positive 10053815 Anti-insulin receptor antibody positive 10053814 Anti-insulin receptor antibody positive 10068226 Application site photosensitivity reaction 10058730 <td>Vaccination site vesicles</td> <td></td> | Vaccination site vesicles | |
| Vascular access site eczema 10085939 Vasculitic rash 10047111 Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 100777117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 1005982 Alveolitis 10061825 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody positive 10053814 Anti-insulin receptor antibody positive 10068226 Application site photosensitivity reaction 10058730 | Vaginal ulceration | 1 1 |
| Vasculitic rash 10047111 Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 <t< td=""><td>Vascular access site dermatitis</td><td>10085938</td></t<> | Vascular access site dermatitis | 10085938 |
| Vernal keratoconjunctivitis 10081000 Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10054929 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin receptor antibody positive 10053814 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthmal late onset 10003553 | Vascular access site eczema | 10085939 |
| Vessel puncture site rash 10077117 Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10061425 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin receptor antibody positive 10053814 Anti-insulin receptor antibody positive 10068226 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthmatic crisis 10064823 Auricula | Vasculitic rash | 10047111 |
| Vessel puncture site vesicles 10077813 Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginal ulceration 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin receptor antibody positive 10053814 Anti-insulin receptor antibody positive 10068226 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 <td>Vernal keratoconjunctivitis</td> <td>L</td> | Vernal keratoconjunctivitis | L |
| Vulval eczema 10066273 Vulval ulceration 10047768 Vulvovaginal rash 10071588 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10054929 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture | Vessel puncture site rash | 10077117 |
| Vulvovaginal rash 10047768 Vulvovaginal rash 10071588 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10053815 Anti-insulin antibody increased 10053815 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthmaic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A incr | Vessel puncture site vesicles | 10077813 |
| Vulvovaginal rash 10071588 Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Anti-ibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Application site photosensitivity reaction 1008225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10005191 Blister 10005191 Blood immunoglobulin A abnormal 10 | Vulval eczema | 10066273 |
| Vulvovaginal ulceration 10050181 Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma 1ate onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005586 | Vulval ulceration | 10047768 |
| Vulvovaginitis allergic 10080783 Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10005191 Blister upture 10073385 Blood immunoglobulin A abnormal 10005586 | Vulvovaginal rash | 10071588 |
| Acute respiratory failure 10001053 Administration site photosensitivity reaction 10075961 Airway remodelling 10075289 Allergy to chemicals 10061626 Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003553 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005586 | Vulvovaginal ulceration | 10050181 |
| Administration site photosensitivity reaction Airway remodelling Allergy to chemicals Allergy to fermented products Alpha tumour necrosis factor increased Alveolitis Antibody test abnormal Antibody test positive Anti-insulin antibody increased Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive Anti-insulin receptor antibody positive Application site photosensitivity reaction Asthma Asthma Asthma late onset Asthma-chronic obstructive pulmonary disease overlap syndrome Asthmatic crisis Auricular swelling Blister Blood immunoglobulin A abnormal Blood immunoglobulin A increased 10061425 10061425 10061425 10061427 10063815 10068226 10068226 10068225 Application site photosensitivity reaction 10078730 10077005 10077005 10077005 10077005 | Vulvovaginitis allergic | 10080783 |
| Alirway remodelling Allergy to chemicals Allergy to fermented products Alpha tumour necrosis factor increased Alveolitis Antibody test abnormal Antibody test positive Anti-insulin antibody increased Anti-insulin antibody positive Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive Anti-insulin receptor antibody positive Application site photosensitivity reaction Asthma Asthma late onset Asthma-chronic obstructive pulmonary disease overlap syndrome Asthmatic crisis Auricular swelling Blister Blood immunoglobulin A abnormal Blood immunoglobulin A increased 10065982 10075289 10075289 10075289 10075289 10075289 10075289 10075289 | Acute respiratory failure | 10001053 |
| Allergy to chemicals Allergy to fermented products 10054929 Alpha tumour necrosis factor increased 10059982 Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10077005 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling Blister 10003594 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005586 | Administration site photosensitivity reaction | 10075961 |
| Allergy to fermented products Alpha tumour necrosis factor increased Alveolitis Antibody test abnormal Antibody test positive Anti-insulin antibody increased Anti-insulin antibody positive Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive Anti-insulin receptor antibody positive Anti-insulin receptor antibody positive Application site photosensitivity reaction Asthma Asthma late onset Asthma-chronic obstructive pulmonary disease overlap syndrome Asthmatic crisis Auricular swelling Blister Blood immunoglobulin A abnormal Blood immunoglobulin A increased 1005586 | Airway remodelling | 10075289 |
| Alpha tumour necrosis factor increased Alveolitis Antibody test abnormal Antibody test positive Anti-insulin antibody increased Anti-insulin antibody positive Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive Anti-insulin receptor antibody positive Application site photosensitivity reaction Asthma Asthma 10003553 Asthma-chronic obstructive pulmonary disease overlap syndrome Asthmatic crisis Auricular swelling Blister Blood immunoglobulin A abnormal Blood immunoglobulin A increased 100018225 10068226 10068225 10068225 10077005 10077005 10077005 10077005 10077005 | Allergy to chemicals | 10061626 |
| Alveolitis 10001889 Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10068226 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 100073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Allergy to fermented products | 10054929 |
| Antibody test abnormal 10061425 Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10068226 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005586 | Alpha tumour necrosis factor increased | 10059982 |
| Antibody test positive 10061427 Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Alveolitis | 10001889 |
| Anti-insulin antibody increased 10053815 Anti-insulin antibody positive 10068226 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005586 | Antibody test abnormal | 10061425 |
| Anti-insulin antibody positive 10053814 Anti-insulin receptor antibody increased 10068226 Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Antibody test positive | 10061427 |
| Anti-insulin receptor antibody increased Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Anti-insulin antibody increased | 10053815 |
| Anti-insulin receptor antibody positive 10068225 Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Anti-insulin antibody positive | 10053814 |
| Application site photosensitivity reaction 10058730 Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Anti-insulin receptor antibody increased | 10068226 |
| Asthma 10003553 Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Anti-insulin receptor antibody positive | 10068225 |
| Asthma late onset 10003559 Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Application site photosensitivity reaction | 10058730 |
| Asthma-chronic obstructive pulmonary disease overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Asthma | 10003553 |
| overlap syndrome 10077005 Asthmatic crisis 10064823 Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Asthma late onset | 10003559 |
| Auricular swelling 10003800 Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | | 10077005 |
| Blister 10005191 Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Asthmatic crisis | 10064823 |
| Blister rupture 10073385 Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Auricular swelling | 10003800 |
| Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Blister | 10005191 |
| Blood immunoglobulin A abnormal 10005584 Blood immunoglobulin A increased 10005586 | Blister rupture | 10073385 |
| Blood immunoglobulin A increased 10005586 | Blood immunoglobulin A abnormal | 10005584 |
| Blood immunoglobulin D increased 10063244 | | 10005586 |
| | Blood immunoglobulin D increased | 10063244 |

| Blood immunoglobulin G abnormal | 10005594 |
|----------------------------------|-----------|
| | 10005596 |
| Blood immunoglobulin G increased | 10005599 |
| Blood immunoglobulin M abnormal | 100055601 |
| Blood immunoglobulin M increased | |
| Bronchial hyperreactivity | 10066091 |
| Bronchial oedema | 10056695 |
| Bullous impetigo | 10006563 |
| Caffeine allergy | 10074895 |
| Capillaritis | 10068406 |
| Charcot-Leyden crystals | 10008413 |
| Cheilitis | 10008417 |
| Childhood asthma | 10081274 |
| Choking | 10008589 |
| Choking sensation | 10008590 |
| Complement factor C1 decreased | 10051552 |
| Complement factor C2 decreased | 10051555 |
| Complement factor C3 decreased | 10050981 |
| Complement factor C4 decreased | 10050983 |
| Complement factor decreased | 10061048 |
| Conjunctivitis | 10010741 |
| Corneal exfoliation | 10064489 |
| Cough variant asthma | 10063076 |
| Cytokine increased | 10085573 |
| Cytokine release syndrome | 10052015 |
| Cytokine storm | 10050685 |
| Ear swelling | 10014025 |
| Eosinophil count abnormal | 10061125 |
| Eosinophil count increased | 10014945 |
| Eosinophil percentage abnormal | 10058133 |
| Eosinophil percentage increased | 10052222 |
| Eosinophilia | 10014950 |
| Eosinophilia myalgia syndrome | 10014952 |
| Eosinophilic bronchitis | 10065563 |
| Eosinophilic oesophagitis | 10064212 |
| Eosinophilic pneumonia | 10014962 |
| Eosinophilic pneumonia acute | 10052832 |
| Eosinophilic pneumonia chronic | 10052833 |
| Erythema | 10015150 |
| Flushing | 10016825 |
| Foreskin oedema | 10085613 |
| Gastrointestinal oedema | 10058061 |

| Generalised oedema 10018092 Genital rash 10018175 Genital swelling 10067639 Haemolytic transfusion reaction 10067122 HLA marker study positive 10082107 Human anti-hamster antibody increased 10082109 Immune complex level increased 10064650 Immunoglobulins abnormal 10021500 Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site panniculitis 10083040 Injection site photosensitivity reaction 1005396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 100448961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 | | • |
|---|---|---|
| Genital swelling 10067639 Haemolytic transfusion reaction 10067122 HLA marker study positive 10067937 Human anti-hamster antibody increased 10082107 Human anti-hamster antibody positive 10082109 Immune complex level increased 10064650 Immunoglobulins abnormal 10021497 Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increas | Generalised oedema | 10018092 |
| Haemolytic transfusion reaction 10067122 HLA marker study positive 10067937 Human anti-hamster antibody increased 10082107 Human anti-hamster antibody positive 10082109 Immune complex level increased 10064650 Immunoglobulins abnormal 10021497 Immunoglobulins increased 10021500 Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site panniculitis 10083040 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 1008773 Medical device site photosensitivity reaction 10076137 Medical device site photosensitivity reaction 100763031 Monocyte chemotactic protein-2 increased 10083043 Mucosal erosion 10028034 Mucosal erosion 10028034 Mucosal erosion 10064486 Mucosal necrosis 10067993 Mucosal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 Noninfective conjunctivitis 10064982 | Genital rash | 10018175 |
| HLA marker study positive 10067937 Human anti-hamster antibody increased 10082107 Human anti-hamster antibody positive 10082109 Immune complex level increased 10064650 Immunoglobulins abnormal 10021497 Immunoglobulins increased 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mucosa vesicle 1002804 Mucosa vesicle 1002803 Mucosal erosion 10064886 Mucosal erosion 10064881 Necrotising panniculitis 1006393 Mucosal erosion 10064993 Mucosal erosion 10062879 Mucosal erosion 10062879 Mucosal oleration 10028034 Necrotising panniculitis 10062579 Neurodermatitis 10064980 Noninfective conjunctivitis 10064982 Noninfective conjunctivitis 10064980 Noninfective conjunctivitis 10064982 | Genital swelling | 10067639 |
| Human anti-hamster antibody increased 10082107 | Haemolytic transfusion reaction | 10067122 |
| Human anti-hamster antibody positive 10082109 | HLA marker study positive | 10067937 |
| Immune complex level increased 10064650 Immunoglobulins abnormal 10021497 Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10044663 Lip exfoliation 10064463 Lip exfoliation 10048961 Macrophage inflammatory protein-1 alpha increased 10048961 Macrophage inflammatory protein-1 alpha increased 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10076331 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosal vesicle 10028034 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10064980 Neurodermatitis 10062579 | Human anti-hamster antibody increased | 10082107 |
| Immunoglobulins abnormal 10021497 Immunoglobulins increased 10021500 Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10048961 Macrophage inflammatory protein-1 alpha increased 10048961 Macrophage inflammatory protein-1 alpha increased 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10076331 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosal vesicle 10028034 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10064980 Neurodermatitis 10062579 Neurodermatitis 10064980 < | Human anti-hamster antibody positive | 10082109 |
| Immunoglobulins increased 10021500 Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site photosensitivity reaction 10083040 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064462 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosa vesicle 10028034 Mucosal erosion 10061297 Mucosal exfoliation 10064980 Mucosal ulceration 10064981 Neutralising antibodies positive 10064980 | Immune complex level increased | 10064650 |
| Immunology test abnormal 10061214 Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site photosensitivity reaction 10083040 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Much ulceration 10028034 Mucosal erosion 10028034 Mucosal erosion 10028034 Mucosal exfoliation 10061297 Mucosal ulceration 10064986 Neurodermatitis 10062579 Neurodermatitis 10064980 < | Immunoglobulins abnormal | 10021497 |
| Implant site photosensitivity 10073415 Infusion site photosensitivity reaction 10065486 Injection site panniculitis 10083040 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosal vesicle 10028034 Mucosal erosion 10061297 Mucosal erosion 10061297 Mucosal ulceration 10064486 Mucosal ulceration 10028124 Nasal crease 10078581 Neurodermatitis 10062579 Neurodermatitis | Immunoglobulins increased | 10021500 |
| Infusion site photosensitivity reaction Injection site panniculitis Injection site photosensitivity reaction Injection site photosensitivity reaction Interstitial lung disease Interstitial lung diseas | Immunology test abnormal | 10061214 |
| Injection site panniculitis 10083040 Injection site photosensitivity reaction 10053396 Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10068773 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028034 Mucosal vesicle 10028103 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Implant site photosensitivity | 10073415 |
| Injection site photosensitivity reaction Interstitial lung disease Inters | Infusion site photosensitivity reaction | 10065486 |
| Interstitial lung disease 10022611 Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Much ulceration 10028034 Mucosal vesicle 10028034 Mucosal erosion 10028084 Mucosal erosion 10061297 Mucosal necrosis 10064980 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Injection site panniculitis | 10083040 |
| Laryngeal dyspnoea 10052390 Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Much ulceration 10028034 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10064486 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Injection site photosensitivity reaction | 10053396 |
| Laryngeal obstruction 10059639 Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosal vesicle 10028084 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10064486 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10029263 Neutralising antibodies positive 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Interstitial lung disease | 10022611 |
| Leukotriene increased 10064663 Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosal vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10064486 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Laryngeal dyspnoea | 10052390 |
| Lip exfoliation 10064482 Localised oedema 10048961 Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucosal vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10064486 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Laryngeal obstruction | 10059639 |
| Localised oedema 10048961 | Leukotriene increased | 10064663 |
| Macrophage inflammatory protein-1 alpha increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10029263 Neurodermatitis 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Lip exfoliation | 10064482 |
| increased 10083049 Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal ulceration 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10062579 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Localised oedema | 10048961 |
| Mechanical urticaria 10068773 Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10062579 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10074701 Non-neutralising antibodies positive 10064982 | Macrophage inflammatory protein-1 alpha | |
| Medical device site photosensitivity reaction 10076137 Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | | |
| Mesenteric panniculitis 10063031 Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | | |
| Monocyte chemotactic protein-2 increased 10083043 Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Medical device site photosensitivity reaction | |
| Mouth ulceration 10028034 Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Mesenteric panniculitis | 10063031 |
| Mucocutaneous ulceration 10028084 Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Monocyte chemotactic protein-2 increased | 10083043 |
| Mucosa vesicle 10028103 Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10064982 | Mouth ulceration | 10028034 |
| Mucosal erosion 10061297 Mucosal exfoliation 10064486 Mucosal necrosis 10067993 Mucosal ulceration 10028124 Nasal crease 10078581 Necrotising panniculitis 10062579 Neurodermatitis 10029263 Neutralising antibodies positive 10064980 Non-neutralising antibodies positive 10074701 Non-neutralising antibodies positive 10064982 | Mucocutaneous ulceration | 10028084 |
| Mucosal exfoliation10064486Mucosal necrosis10067993Mucosal ulceration10028124Nasal crease10078581Necrotising panniculitis10062579Neurodermatitis10029263Neutralising antibodies positive10064980Noninfective conjunctivitis10074701Non-neutralising antibodies positive10064982 | Mucosa vesicle | 10028103 |
| Mucosal necrosis10067993Mucosal ulceration10028124Nasal crease10078581Necrotising panniculitis10062579Neurodermatitis10029263Neutralising antibodies positive10064980Noninfective conjunctivitis10074701Non-neutralising antibodies positive10064982 | Mucosal erosion | |
| Mucosal ulceration10028124Nasal crease10078581Necrotising panniculitis10062579Neurodermatitis10029263Neutralising antibodies positive10064980Noninfective conjunctivitis10074701Non-neutralising antibodies positive10064982 | Mucosal exfoliation | 10064486 |
| Nasal crease10078581Necrotising panniculitis10062579Neurodermatitis10029263Neutralising antibodies positive10064980Noninfective conjunctivitis10074701Non-neutralising antibodies positive10064982 | Mucosal necrosis | 10067993 |
| Necrotising panniculitis10062579Neurodermatitis10029263Neutralising antibodies positive10064980Noninfective conjunctivitis10074701Non-neutralising antibodies positive10064982 | Mucosal ulceration | 10028124 |
| Neurodermatitis10029263Neutralising antibodies positive10064980Noninfective conjunctivitis10074701Non-neutralising antibodies positive10064982 | Nasal crease | 10078581 |
| Neutralising antibodies positive 10064980 Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Necrotising panniculitis | 10062579 |
| Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Neurodermatitis | 10029263 |
| Noninfective conjunctivitis 10074701 Non-neutralising antibodies positive 10064982 | Neutralising antibodies positive | 10064980 |
| Non-neutralising antibodies positive 10064982 | | 10074701 |
| Occupational asthma 10070836 | | 10064982 |
| | Occupational asthma | 10070836 |

| Occupational dermatities | 10030012 |
|----------------------------------------|----------|
| Occupational dermatitis Oedema mucosal | 10030012 |
| | 10030111 |
| Oral mucosal exfoliation | 10004487 |
| Orbital oedema | 10031031 |
| Panniculitis | |
| Penile exfoliation | 10064485 |
| Penile oedema | 10066774 |
| Penile rash | 10082571 |
| Penile swelling | 10034319 |
| Perineal rash | 10075364 |
| Perivascular dermatitis | 10064986 |
| Photosensitivity reaction | 10034972 |
| Pneumonitis | 10035742 |
| Prurigo | 10037083 |
| Pruritus | 10037087 |
| Pulmonary eosinophilia | 10037382 |
| Reactive airways dysfunction syndrome | 10070832 |
| Respiratory arrest | 10038669 |
| Respiratory distress | 10038687 |
| Respiratory failure | 10038695 |
| Respiratory tract oedema | 10070774 |
| Reversible airways obstruction | 10062109 |
| Rhinitis perennial | 10039094 |
| Scrotal exfoliation | 10081178 |
| Scrotal swelling | 10039759 |
| Seasonal allergy | 10048908 |
| Septal panniculitis | 10056876 |
| Skin erosion | 10040840 |
| Skin exfoliation | 10040844 |
| Skin oedema | 10058679 |
| Skin swelling | 10053262 |
| Sneezing | 10041232 |
| Status asthmaticus | 10041961 |
| Stomatitis | 10042128 |
| Streptokinase antibody increased | 10053797 |
| Stridor | 10042241 |
| Suffocation feeling | 10042444 |
| Sunscreen sensitivity | 10083629 |
| Throat tightness | 10043528 |
| Tongue exfoliation | 10064488 |
| Tracheal obstruction | 10044291 |
| | L |

#### Statistical Analysis Plan for Final Analysis Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

#### Mitsubishi Tanabe Pharma Corporation

| Tracheostomy | 10044320 |
|-------------------------------------------------|----------|
| Transplantation associated food allergy | 10075008 |
| Upper airway obstruction | 10067775 |
| Vaccination site photosensitivity reaction | 10076186 |
| Vaccine associated enhanced disease | 10085491 |
| Vaccine associated enhanced respiratory disease | 10085001 |
| Vaginal oedema | 10063818 |
| Visceral oedema | 10065768 |
| Vulval oedema | 10047763 |
| Vulvovaginal exfoliation | 10083435 |
| Vulvovaginal swelling | 10071211 |
| Wheezing | 10047924 |

### **APPENDIX 4 PIMD**

| PT |
|----------------------------------------------------------|
| Acute cutaneous lupus erythematosus |
| Acute disseminated encephalomyelitis |
| Acute febrile neutrophilic dermatosis |
| Acute flaccid myelitis |
| Acute haemorrhagic leukoencephalitis |
| Acute haemorrhagic oedema of infancy |
| Acute macular neuroretinopathy |
| Acute motor axonal neuropathy |
| Acute motor-sensory axonal neuropathy |
| Acute necrotising myelitis |
| Addison's disease |
| Administration site vasculitis |
| Alopecia areata |
| Alveolar proteinosis |
| Ankylosing spondylitis |
| Anti-glomerular basement membrane disease |
| Anti-LRP2 nephropathy |
| Anti-myelin-associated glycoprotein associated |
| polyneuropathy |
| Anti-neutrophil cytoplasmic antibody positive vasculitis |
| Antiphospholipid syndrome |
| Anti-RNA polymerase III antibody increased |
| Anti-RNA polymerase III antibody positive |
| Antisynthetase syndrome |
| Aortitis |
| Application site vasculitis |
| Arteritis |
| Arteritis coronary |
| Arthritis enteropathic |
| Arthritis reactive |
| Atrophic thyroiditis |
| Autoimmune anaemia |
| Autoimmune aplastic anaemia |
| Autoimmune arthritis |
| Autoimmune blistering disease |
| Autoimmune cholangitis |
| Autoimmune colitis |
| Autoimmune demyelinating disease |

| Autoimmune dermatitis |
|---------------------------------------------|
| Autoimmune disorder |
| Autoimmune encephalopathy |
| Autoimmune endocrine disorder |
| Autoimmune enteropathy |
| Autoimmune eye disorder |
| Autoimmune haemolytic anaemia |
| Autoimmune heparin-induced thrombocytopenia |
| Autoimmune hepatitis |
| Autoimmune hyperlipidaemia |
| Autoimmune hypothyroidism |
| Autoimmune inner ear disease |
| Autoimmune lung disease |
| Autoimmune lymphoproliferative syndrome |
| Autoimmune myocarditis |
| Autoimmune myositis |
| Autoimmune nephritis |
| Autoimmune neuropathy |
| Autoimmune neutropenia |
| Autoimmune pancreatitis |
| Autoimmune pancytopenia |
| Autoimmune pericarditis |
| Autoimmune retinopathy |
| Autoimmune thyroid disorder |
| Autoimmune thyroiditis |
| Autoimmune uveitis |
| Autoinflammatory disease |
| Axial spondyloarthritis |
| Axonal and demyelinating polyneuropathy |
| Axonal neuropathy |
| Basedow's disease |
| Behcet's syndrome |
| Bell's palsy |
| Bickerstaff's encephalitis |
| Birdshot chorioretinopathy |
| Brachial plexopathy |
| Bulbar palsy |
| C1q nephropathy |
| Capillaritis |
| Capillary leak syndrome |
| Caplan's syndrome |

| Cardiac sarcoidosis |
|-----------------------------------------------------------|
| Central nervous system lupus |
| Central nervous system vasculitis |
| Cerebral arteritis |
| Cholangitis sclerosing |
| Chronic autoimmune glomerulonephritis |
| Chronic cutaneous lupus erythematosus |
| Chronic inflammatory demyelinating polyradiculoneuropathy |
| Chronic lymphocytic inflammation with pontine |
| perivascular enhancement responsive to steroids |
| Chronic pigmented purpura |
| Clinically isolated syndrome |
| Coeliac disease |
| Cogan's syndrome |
| Cold type haemolytic anaemia |
| Colitis erosive |
| Colitis microscopic |
| Colitis ulcerative |
| Collagen-vascular disease |
| Concentric sclerosis |
| Coombs positive haemolytic anaemia |
| Cranial nerve disorder |
| Cranial nerve palsies multiple |
| Cranial nerve paralysis |
| CREST syndrome |
| Crohn's disease |
| Cutaneous lupus erythematosus |
| Cutaneous sarcoidosis |
| Cutaneous vasculitis |
| Demyelinating polyneuropathy |
| Demyelination |
| Dermatitis bullous |
| Dermatitis barrous Dermatitis herpetiformis |
| Dermatomyositis Diffuse vasculitis |
| Encephalitis allergic |
| Encephalitis autoimmune |
| Encephalitis brain stem |
| Encephalitis haemorrhagic |
| Encephalitis periaxialis diffusa |

| Encephalitis post immunisation Encephalitis toxic Encephalomyelitis Endocrine ophthalmopathy Enteropathic spondylitis Eosinophilic fasciitis Eosinophilic granulomatosis with polyangiitis Erythema induratum Erythema induratum Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis Haemorrhagic vasculitis |
|---|
| Encephalomyelitis Endocrine ophthalmopathy Enteropathic spondylitis Eosinophilic fasciitis Eosinophilic granulomatosis with polyangiitis Erythema induratum Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatous dermatitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Endocrine ophthalmopathy Enteropathic spondylitis Eosinophilic fasciitis Eosinophilic granulomatosis with polyangiitis Erythema induratum Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis rapidly progressive Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Enteropathic spondylitis Eosinophilic fasciitis Eosinophilic granulomatosis with polyangiitis Erythema induratum Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paralysis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Eosinophilic fasciitis Eosinophilic granulomatosis with polyangiitis Erythema induratum Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Eosinophilic granulomatosis with polyangiitis Erythema induratum Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Erythema induratum Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Erythema multiforme Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Erythema nodosum Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Evans syndrome Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Expanded disability status scale score decreased Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Expanded disability status scale score increased Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Facial paralysis Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Facial paresis Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Felty's syndrome Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Fibrillary glomerulonephritis Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Fulminant type 1 diabetes mellitus Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Giant cell arteritis Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Giant cell myocarditis Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Glomerulonephritis membranous Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Glomerulonephritis rapidly progressive Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Glossopharyngeal nerve paralysis Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Goodpasture's syndrome Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Gout Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Gouty arthritis Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Gouty tophus Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Granulomatosis with polyangiitis Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Granulomatous dermatitis Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Guillain-Barre syndrome Haemorrhagic occlusive retinal vasculitis |
| Haemorrhagic occlusive retinal vasculitis |
| Haemorrhagic vasculitis |
| Trachiorinagic vascumus |
| Hashimoto's encephalopathy |
| Hashitoxicosis |
| Henoch-Schonlein purpura |
| Henoch-Schonlein purpura nephritis |
| Hypersensitivity vasculitis |
| Hypoglossal nerve paralysis |
| Hypoglossal nerve paresis |
| Idiopathic inflammatory myopathy |

| Idiopathic interstitial pneumonia |
|---------------------------------------|
| Idiopathic pulmonary fibrosis |
| IgA nephropathy |
| IgM nephropathy |
| IIIrd nerve paralysis |
| IIIrd nerve paresis |
| Immune thrombocytopenia |
| Immune-mediated adrenal insufficiency |
| Immune-mediated adverse reaction |
| Immune-mediated adverse reaction |
| Immune-mediated cholangitis |
| Immune-mediated cholestasis |
| Immune-mediated cystitis |
| Immune-mediated cytopenia |
| Immune-mediated dermatitis |
| Immune-mediated encephalitis |
| Immune-mediated encephalopathy |
| Immune-mediated endocrinopathy |
| Immune-mediated enterocolitis |
| Immune-mediated gastritis |
| Immune-mediated hepatic disorder |
| Immune-mediated hepatitis |
| Immune-mediated hyperthyroidism |
| Immune-mediated hypophysitis |
| Immune-mediated hypothyroidism |
| Immune-mediated lung disease |
| Immune-mediated myocarditis |
| Immune-mediated myositis |
| Immune-mediated nephritis |
| Immune-mediated neurological disorder |
| Immune-mediated neuropathy |
| Immune-mediated oesophagitis |
| Immune-mediated pancreatitis |
| Immune-mediated renal disorder |
| Immune-mediated thyroiditis |
| Immune-mediated uveitis |
| Immunoglobulin G4 related disease |
| Inclusion body myositis |
| Inflammatory bowel disease |
| Injection site vasculitis |
| Insulin autoimmune syndrome |
| IIIoniii uutoiiiiiitalio ojiiatoiiio |

| Interstitial granulomatous dermatitis |
|---------------------------------------------------|
| Interstitial lung disease |
| Intramyelinic oedema |
| IVth nerve paralysis |
| IVth nerve parasis |
| Juvenile idiopathic arthritis |
| Juvenile polymyositis |
| Juvenile porjatic arthritis |
| Juvenile spondyloarthritis Kawasaki's disease |
| Keratoderma blenorrhagica |
| Langerhans' cell histiocytosis |
| Laryngeal rheumatoid arthritis |
| Latent autoimmune diabetes in adults |
| Leukoencephalomyelitis |
| Leukoencephalopathy |
| Lewis-Sumner syndrome |
| Lichen planopilaris |
| Lichen planus |
| Limbic encephalitis |
| Linear IgA disease |
| Liver sarcoidosis |
| Loefgren syndrome |
| Lumbosacral radiculoplexus neuropathy |
| Lupoid hepatic cirrhosis |
| Lupus anticoagulant hypoprothrombinaemia syndrome |
| Lupus cystitis |
| Lupus encephalitis |
| Lupus endocarditis |
| Lupus enteritis |
| Lupus hepatitis |
| Lupus myocarditis |
| Lupus myositis |
| Lupus nephritis |
| Lupus pancreatitis |
| Lupus pleurisy |
| Lupus pneumonitis |
| Lupus vasculitis |
| Lupus-like syndrome |
| Lymphocytic hypophysitis |

| MAGIC syndrome |
|---------------------------------------------------------------------|
| Marburg's variant multiple sclerosis |
| Marine Lenhart syndrome |
| Melkersson-Rosenthal syndrome |
| Membranous-like glomerulopathy with masked |
| IgG-kappa deposits |
| Mesangioproliferative glomerulonephritis |
| Metastatic cutaneous Crohn's disease |
| Microscopic enteritis |
| Microscopic polyangiitis |
| Miller Fisher syndrome |
| Mixed connective tissue disease |
| Mononeuritis |
| Mononeuropathy multiplex |
| Morphoea |
| Multifocal motor neuropathy |
| Multiple sclerosis |
| Multiple sclerosis pseudo relapse |
| Multiple sclerosis relapse |
| Multiple sclerosis relapse prophylaxis |
| Multisystem inflammatory syndrome |
| Multisystem inflammatory syndrome in adults |
| Multisystem inflammatory syndrome in children |
| Muscular sarcoidosis |
| Myasthenia gravis |
| Myasthenia gravis crisis |
| Myasthenic syndrome |
| Myelin oligodendrocyte glycoprotein antibody-<br>associated disease |
| Myelitis |
| Myelitis transverse |
| Myocarditis |
| Narcolepsy |
| Neuralgic amyotrophy |
| Neuritis |
| Neuritis cranial |
| Neuromyelitis optica pseudo relapse |
| Neuromyelitis optica spectrum disorder |
| Neuropsychiatric lupus |
| Neurosarcoidosis |
| Nodular vasculitis |
| INOUUIAF VASCUIIUS |

| Noninfectious myelitis |
|-------------------------------------------------|
| Noninfective encephalitis |
| Noninfective encephalomyelitis |
| Ocular myasthenia |
| Ocular pemphigoid |
| Ocular sarcoidosis |
| Ocular vasculitis |
| Oculofacial paralysis |
| Olfactory nerve disorder |
| Optic ischaemic neuropathy |
| Optic neuritis |
| Optic neuropathy |
| Optic perineuritis |
| Overlap syndrome |
| Palindromic rheumatism |
| Palisaded neutrophilic granulomatous dermatitis |
| Palpable purpura |
| Panencephalitis |
| Paresis cranial nerve |
| Pemphigoid |
| Pemphigus |
| Pericarditis |
| Pericarditis lupus |
| Pericarditis rheumatic |
| Peripheral spondyloarthritis |
| Peritonitis lupus |
| Pernicious anaemia |
| Pleuroparenchymal fibroelastosis |
| Polyarteritis nodosa |
| Polychondritis |
| Polyglandular autoimmune syndrome type I |
| Polyglandular autoimmune syndrome type II |
| Polyglandular autoimmune syndrome type III |
| Polymyalgia rheumatica |
| Polymyositis |
| Polyneuropathy idiopathic progressive |
| Primary biliary cholangitis |
| Primary progressive multiple sclerosis |
| Proctitis ulcerative |
| Progressive facial hemiatrophy |
| Progressive multiple sclerosis |

| Durania alamaia |
|---------------------------------------------------|
| Progressive relapsing multiple sclerosis |
| Psoriasis |
| Psoriatic arthropathy |
| Pulmonary fibrosis |
| Pulmonary renal syndrome |
| Pulmonary sarcoidosis |
| Pulmonary vasculitis |
| Pyoderma gangrenosum |
| Pyostomatitis vegetans |
| Radiculitis brachial |
| Radiologically isolated syndrome |
| Rasmussen encephalitis |
| Raynaud's phenomenon |
| Relapsing multiple sclerosis |
| Relapsing-remitting multiple sclerosis |
| Renal arteritis |
| Renal vasculitis |
| Retinal occlusive vasculitis |
| Retinal vasculitis |
| Reynold's syndrome |
| Rheumatic brain disease |
| Rheumatic disorder |
| Rheumatoid arthritis |
| Rheumatoid arthritis-associated interstitial lung |
| disease |
| Rheumatoid bursitis |
| Rheumatoid lung |
| Rheumatoid meningitis |
| Rheumatoid neutrophilic dermatosis |
| Rheumatoid nodule |
| Rheumatoid scleritis |
| Rheumatoid vasculitis |
| Sarcoidosis |
| Satoyoshi syndrome |
| Sclerodactylia |
| Scleroderma |
| Scleroderma associated digital ulcer |
| Scleroderma renal crisis |
| Secondary progressive multiple sclerosis |
| Segmented hyalinising vasculitis |
| Shrinking lung syndrome |

| Ci14.1 |
|---------------------------------------------------------------|
| Silent thyroiditis |
| Sjogren's syndrome |
| SJS-TEN overlap |
| SLE arthritis |
| Spondylitis |
| Spondyloarthropathy |
| Stevens-Johnson syndrome |
| Still's disease |
| Stoma site vasculitis |
| Subacute cutaneous lupus erythematosus |
| Subacute inflammatory demyelinating polyneuropathy |
| Susac's syndrome |
| Sympathetic ophthalmia |
| Systemic lupus erythematosus |
| Systemic lupus erythematosus disease activity index abnormal |
| Systemic lupus erythematosus disease activity index decreased |
| Systemic lupus erythematosus disease activity index increased |
| Systemic lupus erythematosus rash |
| Systemic scleroderma |
| Systemic sclerosis pulmonary |
| Takayasu's arteritis |
| Terminal ileitis |
| Testicular autoimmunity |
| Thromboangiitis obliterans |
| Thrombocytopenic purpura |
| Thrombosis with thrombocytopenia syndrome |
| Thrombotic thrombocytopenic purpura |
| Tongue paralysis |
| Toxic epidermal necrolysis |
| Trigeminal nerve paresis |
| Trigeminal palsy |
| Tubulointerstitial nephritis and uveitis syndrome |
| Tumefactive multiple sclerosis |
| Type 1 diabetes mellitus |
| Uhthoff's phenomenon |
| Ulcerative keratitis |
| Undifferentiated connective tissue disease |
| Undifferentiated spondyloarthritis |

#### Statistical Analysis Plan for Final Analysis Protocol No. MT-2766-A-101 (CP-PRO-CoVLP-028)

#### Mitsubishi Tanabe Pharma Corporation

| Urticarial vasculitis |
|-------------------------------------------------|
| Uveitis |
| Vaccination site vasculitis |
| Vaccine associated enhanced disease |
| Vaccine associated enhanced respiratory disease |
| Vagus nerve paralysis |
| Vascular purpura |
| Vasculitic rash |
| Vasculitic ulcer |
| Vasculitis |
| Vasculitis gastrointestinal |
| Vasculitis necrotising |
| VIth nerve paralysis |
| VIth nerve paresis |
| Vitiligo |
| Vocal cord paralysis |
| Vocal cord paresis |
| Vogt-Koyanagi-Harada disease |
| Warm type haemolytic anaemia |
| XIth nerve paralysis |